CLINICAL TRIAL: NCT02432274
Title: Phase 1/2 Study of Lenvatinib in Children and Adolescents With Refractory or Relapsed Solid Malignancies and Young Adults With Osteosarcoma
Brief Title: Study of Lenvatinib in Children and Adolescents With Refractory or Relapsed Solid Malignancies and Young Adults With Osteosarcoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Eisai Limited (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Organization: Eisai Inc. (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: E7080-G000-207; 2013-005534-38 (EudraCT Number)
Record Dates: First submitted 2015-04-22; First posted 2015-05-04 (Estimated); Results first posted 2020-09-17 (Actual); Last update posted 2023-07-11 (Actual); Status verified 2021-08

CONDITIONS: Tumors; Solid Malignant Tumors; Osteosarcoma; Differentiated Thyroid Cancer (DTC)
Keywords: E7080; Lenvatinib; Solid malignancies; Osteosarcoma; Differentiated Thyroid Cancer
MeSH Terms: conditions — Neoplasms; Osteosarcoma | interventions — lenvatinib; Ifosfamide; Etoposide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Cohort 1: Single-Agent Dose-Finding (Experimental): Children and adolescents with relapsed or refractory solid malignant tumors.
  Interventions: Drug: Lenvatinib
- Cohort 2A: Single-agent Expansion (DTC) (Experimental): Children and adolescents with 131 iodine-refractory DTC.
  Interventions: Drug: Lenvatinib
- Cohort 2B: Single-agent Expansion (Osteosarcoma) (Experimental): Participants with relapsed or refractory osteosarcoma.
  Interventions: Drug: Lenvatinib
- Cohort 3A: Combination Dose-finding (Experimental): Participants with relapsed or refractory osteosarcoma will receive lenvatinib in combination with ifosfamide and etoposide.
  Interventions: Drug: Lenvatinib; Drug: Ifosfamide; Drug: Etoposide
- Cohort 3B: Combination Expansion (Experimental): Participants with relapsed or refractory osteosarcoma will receive lenvatinib in combination with ifosfamide and etoposide.
  Interventions: Drug: Lenvatinib; Drug: Ifosfamide; Drug: Etoposide

INTERVENTIONS:
Drug: Lenvatinib — Cohort 1: Lenvatinib will be administered orally, once daily on Days 1 to 28 of each 28-day cycle at a starting dose of 11 mg/m2. Dose can be de-escalated to 9 mg/m2 or escalated to 14 and 17 mg/m2.
  Other Names: E7080, lenvatinib
  Arms: Cohort 1: Single-Agent Dose-Finding
Drug: Lenvatinib — Cohort 2A: Lenvatinib (RD determined in Cohort 1) will be administered orally, once daily on Days 1 to 28 of each 28-day cycle.
  Other Names: E7080, lenvatinib
  Arms: Cohort 2A: Single-agent Expansion (DTC)
Drug: Lenvatinib — Cohort 2B: Lenvatinib (RD determined in Cohort 1) will be administered orally, once daily on Days 1 to 28 of each 28-day cycle.
  Other Names: E7080, lenvatinib
  Arms: Cohort 2B: Single-agent Expansion (Osteosarcoma)
Drug: Lenvatinib — Cohort 3A: Lenvatinib will be administered orally, once daily on Days 1 to 21 of each 21-day cycle at 20% lower than RD determined in Cohort 1 (starting dose). Lenvatinib dose can be escalated to the RD from Cohort 1 or de-escalated to 40 and 60% lower than the RD from Cohort 1.
  Other Names: E7080, lenvatinib
  Arms: Cohort 3A: Combination Dose-finding
Drug: Lenvatinib — Cohort 3B: Lenvatinib will be administered orally, once daily on Days 1 to 21 of each 21-day cycle at the RD as determined in Cohort 3A.
  Other Names: E7080, lenvatinib
  Arms: Cohort 3B: Combination Expansion
Drug: Ifosfamide — Ifosfamide 3000 mg/m2/day (starting dose) will be administered on Days 1 to 3 of each 21-day cycle for a total of 5 cycles. Ifosfamide dose can be de-escalated to 2400 mg/m2/day and 1800 mg/m2/day.
  Arms: Cohort 3A: Combination Dose-finding
Drug: Etoposide — Etoposide 100 mg/m2/day (starting dose) will be administered on Days 1 to 3 of each 21-day cycle for a total of 5 cycles. Etoposide dose can be de-escalated to 80 mg/m2/day and 60 mg/m2/day.
  Arms: Cohort 3A: Combination Dose-finding
Drug: Ifosfamide — Ifosfamide dose identified in Cohort 3A will be administered on Days 1 to 3 of each 21-day cycle for a total of 5 cycles.
  Arms: Cohort 3B: Combination Expansion
Drug: Etoposide — Etoposide dose identified in Cohort 3A will be administered on Days 1 to 3 of each 21-day cycle for a total of 5 cycles.
  Arms: Cohort 3B: Combination Expansion

SUMMARY:
This is a phase 1/2 study evaluating safety, tolerability, and efficacy of lenvatinib as single-agent, and in combination with chemotherapy (ifosfamide and etoposide) in children and adolescents with refractory or relapsed solid malignancies including differentiated thyroid carcinoma (single agent lenvatinib) and osteosarcoma (single agent and combination lenvatinib).

DETAILED DESCRIPTION:
The study consists of 5 cohorts:

Cohort 1 (Single-Agent Dose-Finding) dose-escalation to find the recommended dose (RD) of lenvatinib using time-to-event continual reassessment method (TiTE-CRM) in children and adolescents with relapsed or refractory solid malignant tumors. When the RD is identified, Cohorts 2A, 2B, and 3A will enroll in parallel.

Cohort 2 (Single-Agent Expansion) will evaluate the efficacy of lenvatinib at the RD in children, adolescents, and young adults with

1. 131 iodine-refractory differentiated thyroid cancer (DTC) [Cohort 2A] or
2. Relapsed or refractory osteosarcoma [Cohort 2B]

Cohort 3A (Combination Dose-Finding) will determine the RD of lenvatinib in combination with ifosfamide and etoposide in children, adolescents, and young adults with relapsed or refractory osteosarcoma.

Cohort 3B (Combination Expansion) will evaluate the efficacy of lenvatinib at the RD from Cohort 3A in combination with ifosfamide and etoposide in children, adolescents, and young adults with relapsed or refractory osteosarcoma. Participants with osteosarcoma who have enrolled into Cohort 1 or 2B and experienced progressive disease will also be candidates for enrollment in Cohort 3B.

Lenvatinib will be provided as hard capsules containing 1, 4, or 10 mg lenvatinib. Lenvatinib capsules should be dissolved in water or apple juice for those who are unable to swallow capsules.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed diagnosis of solid malignant tumor.

   1. Cohort 1: Any solid malignant tumor.
   2. Cohort 2A: Differentiated Thyroid Cancer (DTC) with one of the following histological subtypes:

   i) Papillary thyroid cancer (PTC). i.a) Follicular variant. i.b) Other variants (including but not limited to tall cell, columnar cell, cribriform-morular, solid, oxyphil, Warthin's-like, trabecular, tumor with nodular fasciitis-like stroma, Hurthle cell variant of papillary carcinoma, or poorly differentiated carcinomas).

   ii) Follicular thyroid cancer (FTC). ii.a) Hurthle cell. ii.b) Clear cell. ii.c) Insular.

   c) Cohort 2B, 3A, and 3B: Relapsed or refractory osteosarcoma.
2. Relapsed or refractory solid tumor malignancy that has progressed on standard anticancer therapy with no available curative options. (Note: Osteosarcoma participants must be in first or subsequent relapse [greater than or equal to first relapse]). Only the osteosarcoma participants enrolled to Cohorts 3A and 3B must be deemed candidates for ifosfamide and etoposide chemotherapy).
3. Evaluable or measurable disease that meets the following criteria:

   1. Participants must have evaluable or measurable disease based on RECIST 1.1 using computed tomography (CT)/magnetic resonance imaging (MRI).
   2. Lesions that have had external beam radiotherapy (EBRT) or locoregional therapies such as radiofrequency (RF) ablation must have subsequently grown unequivocally to be deemed a target lesion.
4. DTC participants must be 131 iodine-refractory/ relapsed as defined by at least one of the following:

   1. One or more evaluable or measurable lesions that do not demonstrate iodine uptake on any radioiodine scan; or
   2. One or more evaluable or measurable lesions that have progressed based on RECIST 1.1, within 12 months of 131 iodine therapy, despite demonstration of radioiodine avidity at the time of that treatment by pre- or post-treatment scanning. These participants must not be eligible for possible curative surgery; or
   3. Cumulative activity of 131 iodine greater than 400 millicuries (mCi) or 14.8 gigabecquerels (GBq), with the last dose administered at least 6 months prior to study entry.
5. Participants with DTC must be receiving thyroxine suppression therapy and levels of thyroid stimulating hormone (TSH) should not be elevated (TSH should be less than or equal to 5.50 milliunits per liter (mU/L)). When tolerated by the participant, thyroxine dose should be changed to achieve TSH suppression (TSH less than 0.50 mU/L).
6. Participants with known central nervous system (CNS) primary tumors or metastases who have completed brain therapy (such as radiotherapy, stereotactic radiosurgery, or surgical resection) and have remained clinically stable, asymptomatic, and off of steroids for 2 weeks prior to Cycle 1 Day 1 will be eligible.
7. Male or female participants age 2 years to less than18 years and less than or equal to 25 years for osteosarcoma subjects at the time of informed consent.
8. Lansky play score greater than or equal to 50% or Karnofsky Performance Status score greater than or equal to 50%. Use Karnofsky for participants greater than or equal to 16 years of age and Lansky for participants less than 16 years of age.
9. Life expectancy greater than or equal to 3 months.
10. Adequate bone marrow function as evidenced by:

    1. absolute neutrophil count (ANC) greater than or equal to 1.0 x 10^9/L (for Cohorts 3A and 3B leucocyte count greater than or equal to 2 x 10^9/L; participants with bone marrow involvement should have ANC greater than or equal to 0.8 x 10^9/L and leucocyte count greater than or equal to 1 x 10^9/L).
    2. hemoglobin greater than or equal to 8.0 grams/deciliter (g/dL) (a hemoglobin less than 8.0 g/dL is acceptable if it is corrected by growth factor or transfusion before starting lenvatinib).
    3. platelet count greater than or equal to 75 x 10^9/L.
11. Adequate liver function as evidenced by:

    1. bilirubin less than or equal 1.5 times the upper limit of normal (ULN).
    2. alkaline phosphatase, alanine aminotransferase (ALT), and aspartate aminotransferase (AST) less than or equal to 3 times ULN.
12. Adequate renal function as evidenced by:

    a) Serum creatinine based on age/gender as below. If serum creatinine is greater than maximum serum creatinine for age/gender as shown in the table below, then creatinine clearance (or radioisotope glomerular filtration rate [GFR]) must be greater than 70 milliliter/minute/1.73 square meter (mL/min/1.73 m2).

    Maximum Serum Creatinine in milligrams/deciliter (mg/dL) for male:

    i. Age 2 to less than 6 years = 0.8

    ii. Age 6 to less than 10 years = 1.0

    iii. Age 10 to less than 13 years = 1.2

    iv. Age 13 to less than 16 years = 1.5

    v. Age greater than or equal to 16 years = 1.7

    Maximum Serum Creatinine (mg/dL) for Female:

    vi. Age 2 to less than 6 years = 0.8

    vii. Age 6 to less than 10 years = 1.0

    viii. Age 10 to less than 13 years = 1.2

    ix. Age 13 to less than 16 years = 1.4

    x. Age greater than or equal to 16 years = 1.4

    The threshold creatinine values in this Table were derived from the Schwartz formula for estimating glomerular filtration rate using child length and stature data published by the CDC.

    b) Urine dipstick less than 2+ for proteinuria. Participants who have greater than or equal to 2+ proteinuria on dipstick urinalysis should undergo a spot protein-creatinine (P/C) ratio that should be Grade less than 2.

    c) No clinical evidence of nephrotic syndrome.
13. Adequate cardiac function as evidenced by left ventricular ejection fraction (LVEF) greater than or equal to 50%) at baseline as determined by echocardiography.
14. Adequately controlled blood pressure (BP) with or without antihypertensive medications, defined as:

    BP less than 95th percentile for sex, age, and height/length at screening (as per National Heart Lung and Blood Institute guidelines) and no change in antihypertensive medications within 1-week prior to Cycle 1/Day 1. Osteosarcoma subjects 18 to 25 years should have BP ≤150/90 mm Hg at screening and no change in antihypertensive therapy within 1 week prior to Cycle 1/Day 1.
15. Washout of 3 weeks in case of prior chemotherapy, 6 weeks if treatment included nitrosoureas; 4 weeks for definitive radiotherapy, and 2 weeks for palliative radiotherapy; 3 months from high-dose chemotherapy and stem cell rescue; 3 weeks from major surgery. Participants must have recovered from the acute toxic effects of all prior anticancer therapy before enrollment into the study.
16. Written and signed informed consent from the parent(s) or legal representative (guardian) and assent from the minor participant. Written informed consent from subjects ≥18 years.
17. Willing and able to comply with the protocol, scheduled follow-up, and management of toxicity as judged by the Investigator.

    Cohort 3B (Combination Expansion): Osteosarcoma subjects who progressed in Cohorts 1 or 2B and opt to receive combination therapy.
18. Osteosarcoma participants receiving combination therapy of lenvatinib with ifosfamide and etoposide should meet only Inclusion Criteria Numbers 6 through 17 (after progression in Cohort 2B).

Exclusion criteria:

1. Any active infection or infectious illness unless fully recovered prior to dosing.
2. Any medical or other condition that in the opinion of the investigator(s) would preclude the participant's participation in a clinical study.
3. Other organ toxicity due to prior anticancer therapy (investigational agent, chemotherapy, or radiation therapy) except alopecia, and ototoxicity due to cisplatin not already covered in the inclusion/exclusion criteria, which has not recovered to Grade less than 2 per Common Terminology Criteria for Adverse Events (CTCAE) v4.0.
4. Known hypersensitivity to any component of the product (lenvatinib or ingredients).
5. Concurrent administration of any other antitumor therapy.
6. Previous treatment with lenvatinib (except for participants previously enrolled into Cohorts 1 or 2B of this study).
7. Two or more prior vascular endothelial growth factor/vascular endothelial growth factor receptor (VEGF/VEGFR) targeted therapies.
8. Currently receiving any investigational drug or device in another clinical trial or within 30 days preceding informed consent.
9. A clinically significant ECG abnormality, including a marked baseline prolonged QT or QTc interval (eg, a repeated demonstration of a QTc interval greater than 480 msec).
10. Gastrointestinal malabsorption or any other condition that in the opinion of the investigator might affect the absorption of lenvatinib.
11. Gastrointestinal bleeding or active hemoptysis (bright red blood of at least half teaspoon) within 3 weeks prior to the first dose of study drug.
12. Active second malignancy within 2 years prior to enrollment ([in addition to the primary tumor types specified by cohort in Inclusion Criterion Number 1], but not including definitively treated superficial melanoma, in-situ, basal or squamous cell carcinoma of the skin).
13. Previous treatment with ifosfamide and Grade greater than or equal to 3 nephrotoxicity or encephalopathy (Cohorts 3A and 3B).
14. Females who are breastfeeding or pregnant at Screening or Baseline (as documented by a positive beta-human chorionic gonadotropin [ß-hCG] (or human chorionic gonadotropin [hCG]) test with a minimum sensitivity of 25 IU/L or equivalent units of ß-hCG [or hCG]). A separate baseline assessment is required if a negative screening pregnancy test was obtained more than 72 hours before the first dose of study drug.

    Cohort 3B (Combination Expansion): Osteosarcoma participants who progressed in Cohorts 1 or 2B and opt to receive combination therapy.
15. Osteosarcoma participants receiving combination therapy of lenvatinib with ifosfamide and etoposide should meet all the exclusion criteria, with the exception of Criterion Number 6.

Ages: 2 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 117 (Actual)
Dates: Start 2014-12-29 (Actual); Primary Completion 2019-07-18 (Actual); Study Completion 2022-07-20 (Actual)

CONTACTS AND LOCATIONS:
Locations (19):
- Texas Children's Hospital, Houston, Texas, United States
- France (7):
  - CHU Strasbourg - Hopital Hautepierre, Strasbourg, Bas Rhin
  - Centre Oscar Lambret Lille, Lille, Rhone
  - Centre Leon Berard, Lyon, Rhone
  - CHU Nantes - Hopital Mere-Enfant, Nantes
  - Institut Curie - Centre de Lutte Contre le Cancer (CLCC) de Paris, Paris
  - Institut Gustave Roussy, Paris
  - CHU de Toulouse - Hopital des Enfants, Toulouse
- Germany (2):
  - Universitaetsklinikum Muenster, Münster
  - Kinderklinik des Olga hospitals, Stuttgart
- Italy (3):
  - Istituto Ortopedico Rizzoli, Bologna
  - Fondazione IRCCS Istituto Nazionale dei Tumori, Milan
  - Ospedale Pediatrico Bambino Gesu, Roma
- Spain (3):
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Infantil Universitario Nino Jesus, Madrid
  - Hospital Universitario y Politecnico La Fe Hospital La Fe Valencia, Valencia
- United Kingdom (3):
  - Birmingham Children's Hospital, Birmingham
  - University College London Hospital, London
  - Royal Victoria Infirmary, Newcastle

REFERENCES:
- [Derived] Gaspar N, Campbell-Hewson Q, Gallego Melcon S, Locatelli F, Venkatramani R, Hecker-Nolting S, Gambart M, Bautista F, Thebaud E, Aerts I, Morland B, Rossig C, Canete Nieto A, Longhi A, Lervat C, Entz-Werle N, Strauss SJ, Marec-Berard P, Okpara CE, He C, Dutta L, Casanova M. Phase I/II study of single-agent lenvatinib in children and adolescents with refractory or relapsed solid malignancies and young adults with osteosarcoma (ITCC-050)☆. ESMO Open. 2021 Oct;6(5):100250. doi: 10.1016/j.esmoop.2021.100250. Epub 2021 Sep 22. PMID 34562750
- [Derived] Rutkowski P. Antiangiogenic agents combined with systemic chemotherapy in refractory osteosarcoma. Lancet Oncol. 2021 Sep;22(9):1206-1207. doi: 10.1016/S1470-2045(21)00422-8. Epub 2021 Aug 17. No abstract available. PMID 34416160
- [Derived] Gaspar N, Venkatramani R, Hecker-Nolting S, Melcon SG, Locatelli F, Bautista F, Longhi A, Lervat C, Entz-Werle N, Casanova M, Aerts I, Strauss SJ, Thebaud E, Morland B, Nieto AC, Marec-Berard P, Gambart M, Rossig C, Okpara CE, He C, Dutta L, Campbell-Hewson Q. Lenvatinib with etoposide plus ifosfamide in patients with refractory or relapsed osteosarcoma (ITCC-050): a multicentre, open-label, multicohort, phase 1/2 study. Lancet Oncol. 2021 Sep;22(9):1312-1321. doi: 10.1016/S1470-2045(21)00387-9. Epub 2021 Aug 17. PMID 34416158
- [Derived] Hattinger CM, Patrizio MP, Magagnoli F, Luppi S, Serra M. An update on emerging drugs in osteosarcoma: towards tailored therapies? Expert Opin Emerg Drugs. 2019 Sep;24(3):153-171. doi: 10.1080/14728214.2019.1654455. Epub 2019 Aug 14. PMID 31401903

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part at 19 investigative sites in France, Germany, Italy, Spain, United Kingdom and the United States. Total 117 participants were enrolled and screened, of which 20 participants were screen failures and 97 participants received study treatment.
Pre-assignment Details: Prior to entering Cohort 1, some participants aged 2 to less than (<) 6 years underwent a run-in period and received lenvatinib 5 milligram per square meter (mg/m^2) per body surface area (BSA) as capsules or suspension once daily for 21 days.
Groups:
- Cohort 1, Single-agent Dose-finding: Lenvatinib 11 mg/m^2: Participants(age group 2 to<6 years and 6 to<18 years)with relapsed or refractory solid malignant tumors received lenvatinib 11mg/m^2(per BSA, daily dose capped at 24 milligram per day[mg/day])as capsules or suspension(lenvatinib capsules dissolved in water/apple juice for participants who were unable to swallow capsules and given as suspension),orally,once daily on Days 1 to 28 of each treatment cycle until progressive disease(PD),intolerable toxicity,participant noncompliance with safety/efficacy assessments,initiation of another anticancer therapy,voluntary discontinuation by participant at any time,or study termination by sponsor,whichever occurred first. Eligible participants of age group 2 to<6 years first underwent 21days run-in period with lenvatinib 5mg/m^2,once daily before receiving lenvatinib11 mg/m^2 in Cycle1 in Cohort1. Duration of each treatment cycle in Cohort1=28 days.After determining recommended dose(RD)in Cohort1,participants were enrolled in Cohorts 2A,2B and 3A.
- Cohort 1, Single-agent Dose-finding: Lenvatinib 14 mg/m^2: Participants (age group 2 to <6 years and 6 to <18 years) with relapsed or refractory solid malignant tumors received lenvatinib 14 mg/m^2 (per BSA, daily dose capped at 24 mg/day) as capsules or suspension (lenvatinib capsules were dissolved in water or apple juice for participants who were unable to swallow capsules and given as suspension), orally, once daily on Days 1 to 28 of each treatment cycle as a single agent until PD, intolerable toxicity, participant noncompliance with safety or efficacy assessments, initiation of another anticancer therapy, voluntary discontinuation by participant at any time, or study termination by sponsor, whichever occurred first. Eligible participants of age group 2 to <6 years first underwent 21-days run-in period with lenvatinib 5 mg/m^2, once daily before receiving lenvatinib 14 mg/m^2 in Cycle 1 in Cohort 1. Duration of each treatment cycle in Cohort 1=28 days. After determining RD in Cohort 1, participants were enrolled in Cohorts 2A, 2B and 3A.
- Cohort 1, Single-agent Dose-finding: Lenvatinib 17 mg/m^2: Participants (of age group 6 to <18 years) with relapsed or refractory solid malignant tumors received dose of lenvatinib 17 mg/m^2 (administered per BSA, daily dose capped at 24 mg/day) as capsules or suspension (lenvatinib capsules were dissolved in water or apple juice for participants who were unable to swallow capsules and given as suspension), orally, once daily on Days 1 to 28 of each treatment cycle as a single agent until PD, intolerable toxicity, participant noncompliance with safety or efficacy assessments, initiation of another anticancer therapy, voluntary discontinuation by the participant at any time, or study termination by the sponsor, whichever occurred first. Duration of each treatment cycle in Cohort 1=28 days. After determining the RD in Cohort 1, participants were enrolled in Cohorts 2A, 2B and 3A.
- Cohort 2A, Single-agent Expansion, DTC: Lenvatinib 14 mg/m^2: Participants with 131 iodine-refractory differentiated thyroid cancer (DTC) received lenvatinib 14 mg/m^2 (administered per BSA with daily dose capped at 24 mg/day) as capsules or suspension (lenvatinib capsules were dissolved in water or apple juice for participants who were unable to swallow capsules and given as suspension), orally, once daily on Days 1 to 28 of each treatment cycle as a single agent until PD, intolerable toxicity, participant noncompliance with safety or efficacy assessments, initiation of another anticancer therapy, voluntary discontinuation by the participant at any time, or study termination by the sponsor, whichever occurred first. Duration of each treatment cycle in Cohort 2A=28 days.
- Cohort2B,Single-agentExpansion,Osteosarcoma:Lenvatinib14mg/m^2: Participants with relapsed or refractory osteosarcoma received lenvatinib 14 mg/m^2 (administered per BSA with daily dose capped at 24 mg/day) as capsule or suspension (lenvatinib capsules were dissolved in water or apple juice for participants who were unable to swallow capsules and given as suspension), orally, once daily on Days 1 to 28 of each treatment cycle as a single agent until PD, intolerable toxicity, participant noncompliance with safety or efficacy assessments, initiation of another anticancer therapy, voluntary discontinuation by the participant at any time, or study termination by the sponsor, whichever occurred first. Duration of each treatment cycle in Cohort 2B=28 days.
- Cohort 3A, Combination Dose-finding: Lenvatinib 11 mg/m^2: Participants with relapsed or refractory osteosarcoma received lenvatinib 11 mg/m^2 (20 percent [%] lower than the RD from Cohort 1; administered per BSA with daily dose capped at 24 mg/day) as capsules or suspension (lenvatinib capsules were dissolved in water or apple juice for participants who were unable to swallow capsules and given as suspension), orally, once daily on Days 1 to 21 of each treatment cycle in combination with ifosfamide 3000 milligram per square meter per day (mg/m^2/day) intravenously and etoposide 100 mg/m^2/day intravenously on Days 1 to 3 of each treatment cycle for up to a total of 5 cycles as a combination therapy. Duration of each treatment cycle in Cohort 3A=21 days. After determining the RD in Cohort 3A, participants were enrolled in Cohort 3B.
- Cohort 3A, Combination Dose-finding: Lenvatinib 14 mg/m^2: Participants with relapsed or refractory osteosarcoma received lenvatinib 14 mg/m^2 (administrated per BSA with daily dose capped at 24 mg/day) as capsules or suspension (lenvatinib capsules were dissolved in water or apple juice for participants who were unable to swallow capsules and given as suspension), orally, once daily on Days 1 to 21 of each treatment cycle in combination with ifosfamide 3000 mg/m^2/day intravenously and etoposide 100 mg/m^2/day intravenously on Days 1 to 3 of each treatment cycle for up to a total of 5 cycles as a combination therapy. Duration of each treatment cycle in Cohort 3A=21 days. After determining the RD in Cohort 3A, participants were enrolled in Cohort 3B.
- Cohort 3B, Combination Expansion: Lenvatinib 14 mg/m^2: Participants with relapsed or refractory osteosarcoma received lenvatinib 14 mg/m^2 (administrated per BSA with daily dose capped at 24 mg/day) as capsules or suspension (lenvatinib capsules were dissolved in water or apple juice for participants who were unable to swallow capsules and given as suspension), orally, once daily on Days 1 to 21 of each treatment cycle in combination with ifosfamide 3000 mg/m^2/day intravenously and etoposide 100 mg/m^2/day intravenously on Days 1 to 3 of each treatment cycle for up to a total of 5 cycles as a combination therapy. Duration of each treatment cycle in Cohort 3B=21 days.
Period: Overall Study
Arm/Group | Cohort 1, Single-agent Dose-finding: Lenvatinib 11 mg/m^2 | Cohort 1, Single-agent Dose-finding: Lenvatinib 14 mg/m^2 | Cohort 1, Single-agent Dose-finding: Lenvatinib 17 mg/m^2 | Cohort 2A, Single-agent Expansion, DTC: Lenvatinib 14 mg/m^2 | Cohort2B,Single-agentExpansion,Osteosarcoma:Lenvatinib14mg/m^2 | Cohort 3A, Combination Dose-finding: Lenvatinib 11 mg/m^2 | Cohort 3A, Combination Dose-finding: Lenvatinib 14 mg/m^2 | Cohort 3B, Combination Expansion: Lenvatinib 14 mg/m^2
Started (The Participants Flow module (including deaths in reasons for not completed) presentation is based on full analysis set. (Full analysis set included all enrolled participants who did not fail study screening).) | 3 | 9 | 11 | 1 | 31 | 7 | 15 | 20
Underwent Run-in Period | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Treated (Safety Population) | 5 (2 participants assigned to lenvatinib17mg/m^2 actually received 11mg/m^2 (dose capped at 24 mg/day).) | 11 (2 participants assigned to lenvatinib17mg/m^2 actually received 14mg/m^2 (dose capped at 24 mg/day).) | 7 | 1 | 31 | 11 (4 participants assigned to lenvatinib14mg/m^2 actually received 11mg/m^2 (dose capped at 24 mg/day).) | 11 | 20
Completed | 1 | 3 | 4 | 1 | 2 | 0 | 5 | 4
Not Completed | 2 | 6 | 7 | 0 | 29 | 7 | 10 | 16
Not completed — Death | 2 | 6 | 7 | 0 | 27 | 7 | 9 | 14
Not completed — Withdrawal of Consent | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 2

BASELINE CHARACTERISTICS:
Population: Full analysis set included all enrolled participants who did not fail study screening.
Groups:
- Cohort 1, Single-agent Dose-finding: Lenvatinib 11 mg/m^2: Participants (age group 2 to <6 years and 6 to <18 years) with relapsed or refractory solid malignant tumors received lenvatinib 11 mg/m^2 (per BSA, daily dose capped at 24 mg/day) as capsules or suspension (lenvatinib capsules were dissolved in water or apple juice for participants who were unable to swallow capsules and given as suspension), orally, once daily on Days 1 to 28 of each treatment cycle as single agent until PD, intolerable toxicity, participant noncompliance with safety or efficacy assessments, initiation of another anticancer therapy, voluntary discontinuation by participant at any time, or study termination by sponsor, whichever occurred first. Eligible participants of age group 2 to <6 years first underwent 21-days run-in period with lenvatinib 5 mg/m^2, once daily before receiving lenvatinib 11 mg/m^2 in Cycle 1 in Cohort 1. Duration of each treatment cycle in Cohort 1=28 days. After determining RD in Cohort 1, participants were enrolled in Cohorts 2A, 2B and 3A.
- Cohort 2A, Single-agent Expansion, DTC: Lenvatinib 14 mg/m^2: Participants with 131 iodine-refractory DTC received lenvatinib 14 mg/m^2 (administered per BSA with daily dose capped at 24 mg/day) as capsules or suspension (lenvatinib capsules were dissolved in water or apple juice for participants who were unable to swallow capsules and given as suspension), orally, once daily on Days 1 to 28 of each treatment cycle as a single agent until PD, intolerable toxicity, participant noncompliance with safety or efficacy assessments, initiation of another anticancer therapy, voluntary discontinuation by the participant at any time, or study termination by the sponsor, whichever occurred first. Duration of each treatment cycle in Cohort 2A=28 days.
- Cohort 3A, Combination Dose-finding: Lenvatinib 11 mg/m^2: Participants with relapsed or refractory osteosarcoma received lenvatinib 11 mg/m^2 (20% lower than the RD from Cohort 1; administered per BSA with daily dose capped at 24 mg/day) as capsules or suspension (lenvatinib capsules were dissolved in water or apple juice for participants who were unable to swallow capsules and given as suspension), orally, once daily on Days 1 to 21 of each treatment cycle in combination with ifosfamide 3000 mg/m^2/day intravenously and etoposide 100 mg/m^2/day intravenously on Days 1 to 3 of each treatment cycle for up to a total of 5 cycles as a combination therapy. Duration of each treatment cycle in Cohort 3A=21 days. After determining the RD in Cohort 3A, participants were enrolled in Cohort 3B.
- Total: Total of all reporting groups
Arm/Group | Cohort 1, Single-agent Dose-finding: Lenvatinib 11 mg/m^2 | Cohort 1, Single-agent Dose-finding: Lenvatinib 14 mg/m^2 | Cohort 1, Single-agent Dose-finding: Lenvatinib 17 mg/m^2 | Cohort 2A, Single-agent Expansion, DTC: Lenvatinib 14 mg/m^2 | Cohort2B,Single-agentExpansion,Osteosarcoma:Lenvatinib14mg/m^2 | Cohort 3A, Combination Dose-finding: Lenvatinib 11 mg/m^2 | Cohort 3A, Combination Dose-finding: Lenvatinib 14 mg/m^2 | Cohort 3B, Combination Expansion: Lenvatinib 14 mg/m^2 | Total
Number analyzed (Participants) | 3 | 9 | 11 | 1 | 31 | 7 | 15 | 20 | 97
Age, Customized [Count of Participants; unit: Participants]
  2 to <6 years | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 3
  6 to <18 years | 2 | 8 | 11 | 1 | 24 | 5 | 11 | 15 | 77
  18 to <=25 years | 0 | 0 | 0 | 0 | 7 | 2 | 3 | 5 | 17
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 5 | 5 | 0 | 18 | 2 | 5 | 7 | 43
  Male | 2 | 4 | 6 | 1 | 13 | 5 | 10 | 13 | 54
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2 | 0 | 4 | 1 | 4 | 3 | 16
  Not Hispanic or Latino | 1 | 4 | 4 | 0 | 15 | 5 | 8 | 10 | 47
  Unknown or Not Reported | 1 | 4 | 5 | 1 | 12 | 1 | 3 | 7 | 34
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 2 | 5 | 3 | 1 | 20 | 6 | 14 | 13 | 64
  More than one race | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 3 | 6
  Unknown or Not Reported | 1 | 4 | 7 | 0 | 9 | 1 | 1 | 4 | 27

OUTCOME MEASURES:

1. Primary Outcome: Cohort 1: Recommended Dose (RD) of Lenvatinib
Description: RD was defined as the dose that had a dose limiting toxicity (DLT) rate closest to the targeted 20% rate. DLT was an adverse drug reaction and was assessed according to common terminology criteria for adverse events (CTCAE) version (v) 4.03 defined as 1) Grade 4 neutropenia for greater than or equal to (>=) 7 days, 2) Grade >=3 thrombocytopenia with bleeding, or lasting greater than (>) 7 days, 3) Grade >=3 febrile neutropenia, 4) Next course of chemotherapy delayed for >=7 days, 5) Grade >=3 non-hematologic toxicity persisting >7 days optimal supportive care, 6) Grade 4 hypertension, confirmed systolic or diastolic blood pressure >25 millimeters of mercury (mmHg) above the 95th percentile for age, or an elevated diastolic blood pressure (that is, >95th percentile for age) not controlled by a single antihypertensive medication within 14 days of use, 7) Grade 3 proteinuria, 8) Any recurrent Grade 2 non-hematological toxicity requiring >=2 interruption and dose reductions.
Time Frame: Cycle 1 (28 days)
Population: Safety analysis set included all participants who received any study drug and had at least one post-baseline safety evaluation.
Measure: Number; unit: milligram per square meter (mg/m^2)
Groups:
- Cohort 1: All Participants: Participants (of age group 2 to <6 years [following the completion of run-in period] and 6 to <18 years) with relapsed or refractory solid malignant tumors received dose of lenvatinib 11 mg/m^2, 14 mg/m^2 or 17 mg/m^2 (administered per BSA, daily dose capped at 24 mg/day) as capsules or suspension (lenvatinib capsules were dissolved in water or apple juice for participants who were unable to swallow capsules and given as suspension), orally, once daily on Days 1 to 28 of each treatment cycle as a single agent until PD, intolerable toxicity, participant noncompliance with safety or efficacy assessments, initiation of another anticancer therapy, voluntary discontinuation by the participant at any time, or study termination by the sponsor, whichever occurred first. Duration of each treatment cycle in Cohort 1=28 days.
Arm/Group | Cohort 1: All Participants
Number analyzed (Participants) | 23
milligram per square meter (mg/m^2) | 14

2. Primary Outcome: Cohort 2A: Number of Participants With Objective Response (OR) of Complete Response (CR) or Partial Response (PR)
Description: OR was defined as participants with best overall response (BOR) of CR or PR as assessed by investigator based on response evaluation criteria in solid tumors (RECIST) version (v) 1.1. For OR, the BOR was defined as the best response (CR or PR for >4 weeks) recorded from the start of the treatment until PD or death whichever occurred first. CR was defined as the disappearance of all target and non-target lesions (non-lymph nodes). All pathological lymph nodes (whether target or non-target) must have a reduction in their short axis <10 millimeters (mm). PR was defined as at least a 30% decrease in the sum of diameter (SOD) of target lesions, taking as reference the baseline sum diameters. PD was defined as at least 20% increase (including an absolute increase of at least 5 mm) in the SOD of target lesions, taking as reference the smallest sum and/or unequivocal progression of existing non-target lesions and/or appearance of 1 or more new lesions.
Time Frame: From date of first dose of study drug until first documentation of PD or death, whichever occurred first (until the data cut-off date, 31 May 2019)
Population: Full analysis set included all enrolled participants who did not fail study screening.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 2A, Single-agent Expansion, DTC: Lenvatinib 14 mg/m^2
Number analyzed (Participants) | 1
Participants | 1

3. Primary Outcome: Cohort 2A: Number of Participants With Best Overall Response (BOR)
Description: BOR was defined as the best response of CR or PR for >4 weeks or SD for >=7 weeks recorded from the start of the treatment until PD or death, whichever occurred first based on RECIST v1.1. CR: disappearance of all target and non-target lesions (non-lymph nodes). All pathological lymph nodes (whether target or non-target) must have a reduction in their short axis <10 mm. PR: at least a 30% decrease in the SOD of target lesions, taking as reference the baseline sum diameters. SD: neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest SOD. PD was defined as at least 20% increase (including an absolute increase of at least 5 mm) in the SOD of target lesions, taking as reference the smallest sum and/or unequivocal progression of existing non-target lesions and/or appearance of 1 or more new lesions.
Time Frame: From first dose of study drug until PD or death, whichever occurred first (until the data cut-off date, 31 May 2019)
Population: Full analysis set included all enrolled participants who did not fail study screening.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 2A, Single-agent Expansion, DTC: Lenvatinib 14 mg/m^2
Number analyzed (Participants) | 1
Participants
  Complete Response | 0
  Partial Response | 1
  Stable Disease | 0

4. Primary Outcome: Cohorts 2B and 3B: Progression-free Survival (PFS) Rate at Month 4
Description: Progression free survival at Month 4 (PFS-4) rate was defined as the percentage of participants who were alive and without PD at Month 4 after the first dose of study drug, based on RECIST v1.1, using a binomial proportion with corresponding 95% confidence interval (CI). PD: >= 20% increase in sum of diameters of target lesions, reference-smallest sum recorded in study (sum at baseline if that was smallest). Sum of diameters must have absolute increase of >=5 mm. Appearance of >=1 new lesions also considered PD.
Time Frame: At Month 4
Population: PFS-4 evaluable set included all participants treated with study drug for at least 4 months or those who died or radiologically progressed within 4 months after first dose, or received anticancer treatment within 4 months after first dose.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort2B,Single-agentExpansion,Osteosarcoma:Lenvatinib14mg/m^2 | Cohort 3B, Combination Expansion: Lenvatinib 14 mg/m^2
Number analyzed (Participants) | 28 | 15
percentage of participants | 32.1 [15.9 to 52.4] | 66.7 [38.4 to 88.2]

5. Primary Outcome: Cohort 3A: Recommended Dose (RD) of Lenvatinib When Given in Combination With Etoposide and Ifosfamide
Description: RD of lenvatinib when given in combination with ifosfamide and etoposide was defined as dose that resulted in no more than 1 DLT per 6 participants,or hematologic DLT in 1 participant and nonhematologic DLT in another participant per 6 participants,upon repeating same dose level.DLT was adverse drug reaction and assessed per CTCAE v4.03 defined as 1)Grade 4 neutropenia for >=10 days,2)Grade >=3 thrombocytopenia with bleeding,or lasting >=10 days,3)Grade >=3 febrile neutropenia lasting >=7 days,4)Next course of chemotherapy delayed for >=7 days,5)Grade >=3 nonhematologic toxicity persisting >7 days despite optimal supportive care,6)Grade 4 hypertension,confirmed systolic or diastolic blood pressure >25 mmHg above 95th percentile for age,or elevated diastolic blood pressure(>95th percentile for age)not controlled by single antihypertensive medication within 14 days use,7)Grade 3 proteinuria,8)Any recurrent Grade 2 nonhematological toxicity requiring >=2 interruption and dose reductions.
Time Frame: Cycle 1 (21 days)
Population: as for outcome 1
Measure: Number; unit: milligram per square meter (mg/m^2)
Groups:
- Cohort 3A: All Participants: Participants with relapsed or refractory osteosarcoma received lenvatinib 11 mg/m^2 (20% lower than the RD from Cohort 1) or 14 mg/m^2, administered per BSA with daily dose capped at 24 mg/day as capsule or suspension (lenvatinib capsules were dissolved in water or apple juice for participants who were unable to swallow capsules and given as suspension), orally, once daily on Days 1 to 21 of each treatment cycle, in combination with ifosfamide 3000 mg/m^2/day intravenously and etoposide 100 mg/m^2/day intravenously on Days 1 to 3 of each treatment cycle for up to a total of 5 cycles as combination therapy. Duration of each treatment cycle in Cohort 3A=21 days.
Arm/Group | Cohort 3A: All Participants
Number analyzed (Participants) | 22
milligram per square meter (mg/m^2) | 14

6. Secondary Outcome: Cohorts 1, 2B, 3A, and 3B: Number of Participants With Best Overall Response (BOR)
Description: BOR: best response of CR or PR for >4 weeks or SD for >=7 weeks from first dose, recorded from start of treatment until PD or death, whichever occurred first based on RECIST v1.1. CR: disappearance of all target and non-target lesions (non-lymph nodes). All pathological lymph nodes (whether target or non-target) must have reduction in their short axis <10 mm. PR: at least 30% decrease in SOD of target lesions, taking as reference the baseline sum diameters. SD: neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest SOD. PD was defined as: at least 20% increase (including an absolute increase of at least 5 mm) in the SOD of target lesions, taking as reference the smallest sum and/or unequivocal progression of existing non-target lesions and/or appearance of 1 or more new lesions. Not evaluable (NE) means BOR of NE or SD of <7 weeks duration. Unknown means no data were available on the case report form.
Time Frame: From date of first dose of study drug until PD or death, whichever occurred first (Cohort 1, Cohort 2B: until the data cut-off date, 31 May 2019; Cohort 3A, Cohort 3B: until the data cut-off date, 18 July 2019)
Population: Full analysis set included all enrolled participants who did not fail study screening. Here "overall number of participants analyzed" signifies participants who were evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Groups:
- Cohort 1, Single-agent Dose-finding: Lenvatinib 11 mg/m^2: Participants (age group 2 to <6 years [following completion of run-in period] and 6 to <18 years) with relapsed or refractory solid malignant tumors received lenvatinib 11 mg/m^2 (per BSA, daily dose capped at 24 mg/day) as capsules or suspension (lenvatinib capsules were dissolved in water or apple juice for participants who were unable to swallow capsules and given as suspension), orally, once daily on Days 1 to 28 of each treatment cycle as single agent until PD, intolerable toxicity, participant noncompliance with safety or efficacy assessments, initiation of another anticancer therapy, voluntary discontinuation by participant at any time, or study termination by sponsor, whichever occurred first. Duration of each treatment cycle in Cohort 1=28 days.
- Cohort 1, Single-agent Dose-finding: Lenvatinib 14 mg/m^2: Participants (age group 2 to <6 years [following completion of run-in period] and 6 to <18 years) with relapsed or refractory solid malignant tumors received lenvatinib 14 mg/m^2 (per BSA, daily dose capped at 24 mg/day) as capsules or suspension (lenvatinib capsules were dissolved in water or apple juice for participants who were unable to swallow capsules and given as suspension), orally, once daily on Days 1 to 28 of each treatment cycle as a single agent until PD, intolerable toxicity, participant noncompliance with safety or efficacy assessments, initiation of another anticancer therapy, voluntary discontinuation by participant at any time, or study termination by sponsor, whichever occurred first. Duration of each treatment cycle in Cohort 1=28 days.
- Cohort 1, Single-agent Dose-finding: Lenvatinib 17 mg/m^2: Participants (of age group 6 to <18 years) with relapsed or refractory solid malignant tumors received dose of lenvatinib 17 mg/m^2 (administered per BSA, daily dose capped at 24 mg/day) as capsules or suspension (lenvatinib capsules were dissolved in water or apple juice for participants who were unable to swallow capsules and given as suspension), orally, once daily on Days 1 to 28 of each treatment cycle as a single agent until PD, intolerable toxicity, participant noncompliance with safety or efficacy assessments, initiation of another anticancer therapy, voluntary discontinuation by the participant at any time, or study termination by the sponsor, whichever occurred first. Duration of each treatment cycle in Cohort 1=28 days.
- Cohort 3A, Combination Dose-finding: Lenvatinib 11 mg/m^2: Participants with relapsed or refractory osteosarcoma received lenvatinib 11 mg/m^2 (20% lower than the RD from Cohort 1; administered per BSA with daily dose capped at 24 mg/day) as capsules or suspension (lenvatinib capsules were dissolved in water or apple juice for participants who were unable to swallow capsules and given as suspension), orally, once daily on Days 1 to 21 of each treatment cycle in combination with ifosfamide 3000 mg/m^2/day intravenously and etoposide 100 mg/m^2/day intravenously on Days 1 to 3 of each treatment cycle for up to a total of 5 cycles as a combination therapy. Duration of each treatment cycle in Cohort 3A=21 days.
- Cohort 3A, Combination Dose-finding: Lenvatinib 14 mg/m^2: Participants with relapsed or refractory osteosarcoma received lenvatinib 14 mg/m^2 (administrated per BSA with daily dose capped at 24 mg/day) as capsules or suspension (lenvatinib capsules were dissolved in water or apple juice for participants who were unable to swallow capsules and given as suspension), orally, once daily on Days 1 to 21 of each treatment cycle in combination with ifosfamide 3000 mg/m^2/day intravenously and etoposide 100 mg/m^2/day intravenously on Days 1 to 3 of each treatment cycle for up to a total of 5 cycles as a combination therapy. Duration of each treatment cycle in Cohort 3A=21 days.
Arm/Group | Cohort 1, Single-agent Dose-finding: Lenvatinib 11 mg/m^2 | Cohort 1, Single-agent Dose-finding: Lenvatinib 14 mg/m^2 | Cohort 1, Single-agent Dose-finding: Lenvatinib 17 mg/m^2 | Cohort2B,Single-agentExpansion,Osteosarcoma:Lenvatinib14mg/m^2 | Cohort 3A, Combination Dose-finding: Lenvatinib 11 mg/m^2 | Cohort 3A, Combination Dose-finding: Lenvatinib 14 mg/m^2 | Cohort 3B, Combination Expansion: Lenvatinib 14 mg/m^2
Number analyzed (Participants) | 3 | 9 | 10 | 30 | 7 | 14 | 18
Participants
  Complete Response | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Partial Response | 0 | 0 | 0 | 2 | 2 | 0 | 3
  Stable Disease | 2 | 5 | 4 | 13 | 3 | 10 | 9
  Progressive Disease | 1 | 2 | 4 | 12 | 2 | 2 | 4
  Not Evaluable or Unknown | 0 | 2 | 2 | 3 | 0 | 2 | 2

7. Secondary Outcome: Cohorts 1, 2B, 3A, and 3B: Objective Response Rate (ORR)
Description: ORR was defined as the percentage of participants with a BOR of CR or PR for >4 weeks or SD for >=7 weeks as assessed by investigator based on RECIST v1.1, recorded from start of study treatment until PD or death whichever occurred first. CR was defined as the disappearance of all target and non-target lesions (non-lymph nodes). All pathological lymph nodes (whether target or non-target) must have a reduction in their short axis <10 mm. PR was defined as at least a 30% decrease in the SOD of target lesions, taking as reference the baseline sum diameters. 95% CI of the ORR were calculated according to Clopper and Pearson method.
Time Frame: as for outcome 6
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 1, Single-agent Dose-finding: Lenvatinib 11 mg/m^2 | Cohort 1, Single-agent Dose-finding: Lenvatinib 14 mg/m^2 | Cohort 1, Single-agent Dose-finding: Lenvatinib 17 mg/m^2 | Cohort2B,Single-agentExpansion,Osteosarcoma:Lenvatinib14mg/m^2 | Cohort 3A, Combination Dose-finding: Lenvatinib 11 mg/m^2 | Cohort 3A, Combination Dose-finding: Lenvatinib 14 mg/m^2 | Cohort 3B, Combination Expansion: Lenvatinib 14 mg/m^2
Number analyzed (Participants) | 3 | 9 | 10 | 30 | 7 | 14 | 18
percentage of participants | 0 [0.0 to 70.8] | 0 [0.0 to 33.6] | 0 [0.0 to 30.8] | 6.7 [0.8 to 22.1] | 28.6 [3.7 to 71.0] | 0 [0.0 to 23.2] | 16.7 [3.6 to 41.4]

8. Secondary Outcome: Cohorts 1, 2A, 2B, 3A and 3B: Duration of Response (DOR)
Description: DOR was defined as time in months from the first documentation confirmed CR or PR until the first documentation of confirmed PD as assessed by investigator based on RECIST v1.1. CR: disappearance of all target and non-target lesions (non-lymph nodes). All pathological lymph nodes (whether target or non-target) must have a reduction in their short axis <10 mm. PR: at least a 30% decrease in the SOD of target lesions, taking as reference the baseline sum diameters. PD: at least 20% increase (including an absolute increase of at least 5 mm) in the SOD of target lesions, taking as reference the smallest sum and/or unequivocal progression of existing non-target lesions and/or appearance of 1 or more new lesions. 95% CI for the median were calculated according to Brookmeyer and Crowley method.
Time Frame: First documentation of CR/PR until first documentation of PD (Cohort 1, Cohort 2A, Cohort 2B: until the data cut-off date, 31 May 2019; Cohort 3A, Cohort 3B: until the data cut-off date, 18 July 2019)
Population: Full analysis set included all enrolled participants who did not fail study screening. Here "overall number of participants analyzed, N" signifies participants who were evaluable for this measure. Here, "N" for Cohort 1 (Lenvatinib 11, 14, 17 mg/m^2) and Cohort 3A (Lenvatinib 14 mg/m^2) is zero as there were no events of CR or PR in these arms.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort 1, Single-agent Dose-finding: Lenvatinib 11 mg/m^2 | Cohort 1, Single-agent Dose-finding: Lenvatinib 14 mg/m^2 | Cohort 1, Single-agent Dose-finding: Lenvatinib 17 mg/m^2 | Cohort 2A, Single-agent Expansion, DTC: Lenvatinib 14 mg/m^2 | Cohort2B,Single-agentExpansion,Osteosarcoma:Lenvatinib14mg/m^2 | Cohort 3A, Combination Dose-finding: Lenvatinib 11 mg/m^2 | Cohort 3A, Combination Dose-finding: Lenvatinib 14 mg/m^2 | Cohort 3B, Combination Expansion: Lenvatinib 14 mg/m^2
Number analyzed (Participants) | 0 | 0 | 0 | 1 | 2 | 2 | 0 | 3
months |  |  |  | 1.9 [NA to NA] — 95% CI could not be estimated as insufficient number of participants were available for analysis. | 4.6 [NA to NA] — 95% CI could not be estimated as insufficient number of participants were available for analysis. | NA [NA to NA] — Median and 95% CI could not be estimated because all participants were censored from the analysis. |  | NA [NA to NA] — Median and 95% CI could not be estimated because all participants were censored from the analysis.

9. Secondary Outcome: Cohorts 1, 2A, 2B, 3A and 3B: Number of Participants Who Experienced Disease Control
Description: Participants were defined as having disease control if they had a BOR of CR or PR for >4 weeks, or SD (minimum duration from first dose to SD >=7 weeks) or if participants had a BOR of CR or Non-CR/Non-PD (minimum duration from first dose to Non-CR/Non-PD >=7 weeks) per RECIST v1.1, recorded from first dose until PD or death whichever occurred first. CR: disappearance of all target/non-target lesions (non-lymph nodes). All pathological lymph nodes (target/non-target) must have a reduction in their short axis <10 mm. PR: at least a 30% decrease in the SOD of target lesions, taking as reference the baseline sum diameters. SD: neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference smallest SOD. Non-CR/Non-PD: persistence of 1 or more non-target lesions, maintenance of tumor marker level above the normal limits.
Time Frame: From first dose of study drug until PD or death, whichever occurred first (Cohort 1, Cohort 2A, Cohort 2B: until the data cut-off date, 31 May 2019; Cohort 3A, Cohort 3B: until the data cut-off date, 18 July 2019)
Population: Full analysis set included all enrolled participants who did not fail study screening.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1, Single-agent Dose-finding: Lenvatinib 11 mg/m^2 | Cohort 1, Single-agent Dose-finding: Lenvatinib 14 mg/m^2 | Cohort 1, Single-agent Dose-finding: Lenvatinib 17 mg/m^2 | Cohort 2A, Single-agent Expansion, DTC: Lenvatinib 14 mg/m^2 | Cohort2B,Single-agentExpansion,Osteosarcoma:Lenvatinib14mg/m^2 | Cohort 3A, Combination Dose-finding: Lenvatinib 11 mg/m^2 | Cohort 3A, Combination Dose-finding: Lenvatinib 14 mg/m^2 | Cohort 3B, Combination Expansion: Lenvatinib 14 mg/m^2
Number analyzed (Participants) | 3 | 9 | 11 | 1 | 31 | 7 | 15 | 20
Participants | 2 | 5 | 5 | 1 | 16 | 5 | 11 | 14

10. Secondary Outcome: Cohorts 1, 2A, 2B, 3A and 3B: Number of Participants Experienced Clinical Benefit
Description: Participants were defined as having clinical benefit if they had a BOR of CR or PR for >4 weeks or durable SD (lasting >=23 weeks) or if participants had a BOR of CR or durable Non-CR/Non-PD (lasting >=23 weeks) as per RECIST v1.1, recorded from first dose until PD or death whichever occurred first. CR: disappearance of all target/non-target lesions (non-lymph nodes). All pathological lymph nodes (whether target/non-target) must have a reduction in their short axis <10 mm. PR: at least a 30% decrease in the SOD of target lesions, taking as reference the baseline sum diameters. SD: neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest SOD. Non-CR/Non-PD:persistence of 1 or more non-target lesions and maintenance of tumor marker level above the normal limits.
Time Frame: as for outcome 9
Population: Full analysis set included all enrolled participants who did not fail study screening.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1, Single-agent Dose-finding: Lenvatinib 11 mg/m^2 | Cohort 1, Single-agent Dose-finding: Lenvatinib 14 mg/m^2 | Cohort 1, Single-agent Dose-finding: Lenvatinib 17 mg/m^2 | Cohort 2A, Single-agent Expansion, DTC: Lenvatinib 14 mg/m^2 | Cohort2B,Single-agentExpansion,Osteosarcoma:Lenvatinib14mg/m^2 | Cohort 3A, Combination Dose-finding: Lenvatinib 11 mg/m^2 | Cohort 3A, Combination Dose-finding: Lenvatinib 14 mg/m^2 | Cohort 3B, Combination Expansion: Lenvatinib 14 mg/m^2
Number analyzed (Participants) | 3 | 9 | 11 | 1 | 31 | 7 | 15 | 20
Participants | 0 | 3 | 4 | 1 | 7 | 4 | 5 | 8

11. Secondary Outcome: Cohorts 1, 2A, 2B, 3A and 3B: Progression-free Survival (PFS)
Description: PFS was defined as the time (in months) from the date of first dose of study drug to the date of first documentation of PD or date of death, whichever occurred first, based on RECIST v1.1. PD was defined as at least a 20% increase in the SOD of target lesions, taking as reference the baseline SOD of target lesions. 95% CI of median were calculated according to Brookmeyer and Crowley method.
Time Frame: as for outcome 9
Population: Full analysis set included all enrolled participants who did not fail study screening.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort 1, Single-agent Dose-finding: Lenvatinib 11 mg/m^2 | Cohort 1, Single-agent Dose-finding: Lenvatinib 14 mg/m^2 | Cohort 1, Single-agent Dose-finding: Lenvatinib 17 mg/m^2 | Cohort 2A, Single-agent Expansion, DTC: Lenvatinib 14 mg/m^2 | Cohort2B,Single-agentExpansion,Osteosarcoma:Lenvatinib14mg/m^2 | Cohort 3A, Combination Dose-finding: Lenvatinib 11 mg/m^2 | Cohort 3A, Combination Dose-finding: Lenvatinib 14 mg/m^2 | Cohort 3B, Combination Expansion: Lenvatinib 14 mg/m^2
Number analyzed (Participants) | 3 | 9 | 11 | 1 | 31 | 7 | 15 | 20
months | 3.7 [0.5 to 5.0] | 6.3 [0.6 to 10.6] | 5.5 [1.4 to 11.3] | 5.5 [NA to NA] — 95% CI could not be estimated as insufficient number of participants were available for analysis. | 3.0 [1.8 to 5.4] | 7.1 [2.1 to NA] — Upper limit of 95% CI could not be estimated because high number of participants were censored from the analysis. | 12.0 [11.1 to 16.1] | 6.9 [4.2 to NA] — Upper limit of 95% CI could not be estimated because high number of participants were censored from the analysis.

12. Secondary Outcome: Cohorts 1, 2A, 2B, 3A and 3B: Time to Progression (TTP)
Description: TTP was defined as the time from the date of first dose of study drug to the date of first documentation of PD based on RECIST 1.1. PD was defined as at least a 20% increase (including an absolute increase of at least 5 mm) in the SOD of target lesions, taking as reference the baseline SOD of target lesions. 95% CI of median were calculated according to Brookmeyer and Crowley method.
Time Frame: From first dose of study drug until PD (Cohort 1, Cohort 2A, Cohort 2B: until the data cut-off date, 31 May 2019; Cohort 3A, Cohort 3B: until the data cut-off date, 18 July 2019)
Population: Full analysis set included all enrolled participants who did not fail study screening.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort 1, Single-agent Dose-finding: Lenvatinib 11 mg/m^2 | Cohort 1, Single-agent Dose-finding: Lenvatinib 14 mg/m^2 | Cohort 1, Single-agent Dose-finding: Lenvatinib 17 mg/m^2 | Cohort 2A, Single-agent Expansion, DTC: Lenvatinib 14 mg/m^2 | Cohort2B,Single-agentExpansion,Osteosarcoma:Lenvatinib14mg/m^2 | Cohort 3A, Combination Dose-finding: Lenvatinib 11 mg/m^2 | Cohort 3A, Combination Dose-finding: Lenvatinib 14 mg/m^2 | Cohort 3B, Combination Expansion: Lenvatinib 14 mg/m^2
Number analyzed (Participants) | 3 | 9 | 11 | 1 | 31 | 7 | 15 | 20
months | 3.7 [0.5 to 5.0] | 6.3 [0.6 to 10.6] | 5.5 [1.4 to 11.3] | 5.5 [NA to NA] — 95% CI could not be estimated as insufficient number of participants were available for analysis. | 3.0 [1.8 to 5.4] | 7.1 [2.1 to NA] — Upper limit of 95% CI could not be estimated because high number of participants were censored from the analysis. | 12.0 [11.1 to 16.1] | 6.9 [4.2 to NA] — Upper limit of 95% CI could not be estimated because high number of participants were censored from the analysis.

13. Secondary Outcome: Cohorts 1, 2A, 2B, 3A and 3B: Overall Survival (OS)
Description: OS was defined as the time from the date of the first dose of study drug until the date of death from any cause. Participants who are lost to follow-up and those who are alive at the date of data cutoff were censored at the date the participant was last known to be alive (or the data cutoff date). 95% CI of median were calculated according to Brookmeyer and Crowley method.
Time Frame: From first dose of study drug until death (Cohort 1, Cohort 2A, Cohort 2B: until the data cut-off date, 31 May 2019; Cohort 3A, Cohort 3B: until the data cut-off date, 18 July 2019)
Population: Full analysis set included all enrolled participants who did not fail study screening.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort 1, Single-agent Dose-finding: Lenvatinib 11 mg/m^2 | Cohort 1, Single-agent Dose-finding: Lenvatinib 14 mg/m^2 | Cohort 1, Single-agent Dose-finding: Lenvatinib 17 mg/m^2 | Cohort 2A, Single-agent Expansion, DTC: Lenvatinib 14 mg/m^2 | Cohort2B,Single-agentExpansion,Osteosarcoma:Lenvatinib14mg/m^2 | Cohort 3A, Combination Dose-finding: Lenvatinib 11 mg/m^2 | Cohort 3A, Combination Dose-finding: Lenvatinib 14 mg/m^2 | Cohort 3B, Combination Expansion: Lenvatinib 14 mg/m^2
Number analyzed (Participants) | 3 | 9 | 11 | 1 | 31 | 7 | 15 | 20
months | 8.1 [3.8 to NA] — Upper limit of 95% CI could not be estimated due to low number of participants with events. | 7.4 [1.3 to NA] — Upper limit of 95% CI could not be estimated due to low number of participants with events. | 7.7 [2.7 to NA] — Upper limit of 95% CI could not be estimated due to low number of participants with events. | 6.1 [NA to NA] — 95% CI could not be estimated as insufficient number of participants were available for analysis. | 10.0 [5.6 to 12.3] | 13.6 [2.4 to 28.0] | NA [8.8 to NA] — Median and upper limit of 95% CI could not be estimated because high number of participants were censored from the analysis. | NA [7.3 to NA] — Median and upper limit of 95% CI could not be estimated because high number of participants were censored from the analysis.

14. Secondary Outcome: Cohorts 1, 2A, 2B, 3A and 3B: Number of Participants With Treatment-emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs)
Description: Number of participants with TEAEs (serious and non-serious adverse events) and SAEs were reported based on their safety assessments of hematology, clinical chemistry, proximal tibial growth, fecal occult blood, physical examinations, regular measurement of vital signs and electrocardiogram parameter values.
Time Frame: From the date of first dose of study drug up to 30 days after the last dose (up to approximately 7 years)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1, Single-agent Dose-finding: Lenvatinib 11 mg/m^2 | Cohort 1, Single-agent Dose-finding: Lenvatinib 14 mg/m^2 | Cohort 1, Single-agent Dose-finding: Lenvatinib 17 mg/m^2 | Cohort 2A, Single-agent Expansion, DTC: Lenvatinib 14 mg/m^2 | Cohort2B,Single-agentExpansion,Osteosarcoma:Lenvatinib14mg/m^2 | Cohort 3A, Combination Dose-finding: Lenvatinib 11 mg/m^2 | Cohort 3A, Combination Dose-finding: Lenvatinib 14 mg/m^2 | Cohort 3B, Combination Expansion: Lenvatinib 14 mg/m^2
Number analyzed (Participants) | 5 | 11 | 7 | 1 | 31 | 11 | 11 | 20
Participants
  TEAEs | 5 | 11 | 7 | 1 | 29 | 11 | 11 | 20
  SAEs | 3 | 7 | 5 | 1 | 21 | 7 | 9 | 16

15. Secondary Outcome: Cohorts 1, 2A, 2B, 3A, and 3B: Number of Participants With Shift From Baseline to Worst Post Baseline Measurements on Urine DipStick for Proteinuria
Description: An aliquot of the urine samples were collected to analyze protein by dipstick method, microscopic examination (if protein was abnormal). The dipstick test gives results in a semi-quantitative manner and results for urinalysis parameters of urine protein can be read as "negative, Trace, plus (+) 1, +2, +3 and +4" indicating proportional concentrations in the urine sample. The plus sign increases with a higher level of proteins in the urine.
Time Frame: Baseline up to approximately 4 years 7 months
Population: Safety analysis set included all participants who received any study drug and had at least one post-baseline safety evaluation. Here "overall number of participants analyzed" signifies participants who were evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1, Single-agent Dose-finding: Lenvatinib 11 mg/m^2 | Cohort 1, Single-agent Dose-finding: Lenvatinib 14 mg/m^2 | Cohort 1, Single-agent Dose-finding: Lenvatinib 17 mg/m^2 | Cohort 2A, Single-agent Expansion, DTC: Lenvatinib 14 mg/m^2 | Cohort2B,Single-agentExpansion,Osteosarcoma:Lenvatinib14mg/m^2 | Cohort 3A, Combination Dose-finding: Lenvatinib 11 mg/m^2 | Cohort 3A, Combination Dose-finding: Lenvatinib 14 mg/m^2 | Cohort 3B, Combination Expansion: Lenvatinib 14 mg/m^2
Number analyzed (Participants) | 5 | 11 | 7 | 1 | 30 | 11 | 11 | 20
Participants
  Baseline: Trace, Worst Post baseline: Negative | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0
  Baseline: Trace, Worst Post baseline: Trace | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 1
  Baseline: +1, Worst Post baseline: Negative | 2 | 3 | 1 | 0 | 0 | 0 | 0 | 0
  Baseline: +1, Worst Post baseline: +1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Baseline: Negative, Worst Post baseline: Negative | 0 | 1 | 0 | 1 | 4 | 0 | 4 | 2
  Baseline: +2, Worst Post baseline: Negative | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0
  Baseline: +3, Worst Post baseline: Negative | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
  Baseline: +3, Worst Post baseline: +1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
  Baseline: +3, Worst Post baseline: +2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Baseline: +3, Worst Post baseline: Trace | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Baseline: +4, Worst Post baseline: Trace | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Baseline: +4, Worst Post baseline: +1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
  Baseline: Negative, Worst Post baseline: Trace | 0 | 0 | 0 | 0 | 5 | 0 | 1 | 3
  Baseline: Negative, Worst Post baseline: +1 | 0 | 0 | 0 | 0 | 7 | 7 | 1 | 1
  Baseline: Negative, Worst Post baseline: +2 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 6
  Baseline: Negative, Worst Post baseline: +3 | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 2
  Baseline: Trace, Worst Post baseline: +1 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0
  Baseline: Trace, Worst Post baseline: +2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Baseline: Trace, Worst Post baseline: +3 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Baseline: +1, Worst Post baseline: Trace | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Baseline: +1, Worst Post baseline: +2 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 1
  Baseline: +1, Worst Post baseline: +3 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
  Baseline: Negative, Worst Post baseline: +4 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Baseline: +1, Worst Post baseline: +4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

16. Secondary Outcome: Cohorts 1, 2A, 2B, 3A and 3B: Number of Participants With Shift From Baseline to Worst Post Baseline Score in Lansky Performance Play Score
Description: Lansky Performance Play Scale rates a child's activity level for <16 years of age. Scores on scale range from 0 (unresponsive) to 100 ( fully active, normal), where 100=fully active, normal; 90=minor restrictions in physically strenuous activity; 80=active, but tires more quickly; 70=both greater restriction of and less time spent in play activity; 60=up and around, but minimal active play, keeps busy with quieter activities; 50=gets dressed, but lies around much of day, no active play, able to participant in quiet play and activities; 40=mostly in bed, participates in quiet activities; 30=in bed, needs assistance even for quiet play; 20=often sleeping, play entirely limited to very passive activities; 10=no play, does not get out of bed; 0=unresponsive. Higher score indicates more activity and lower indicates less or no activity.
Time Frame: Baseline up to approximately 4 years 7 months
Population: as for outcome 15
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1, Single-agent Dose-finding: Lenvatinib 11 mg/m^2 | Cohort 1, Single-agent Dose-finding: Lenvatinib 14 mg/m^2 | Cohort 1, Single-agent Dose-finding: Lenvatinib 17 mg/m^2 | Cohort 2A, Single-agent Expansion, DTC: Lenvatinib 14 mg/m^2 | Cohort2B,Single-agentExpansion,Osteosarcoma:Lenvatinib14mg/m^2 | Cohort 3A, Combination Dose-finding: Lenvatinib 11 mg/m^2 | Cohort 3A, Combination Dose-finding: Lenvatinib 14 mg/m^2 | Cohort 3B, Combination Expansion: Lenvatinib 14 mg/m^2
Number analyzed (Participants) | 3 | 7 | 7 | 1 | 15 | 6 | 7 | 9
Participants
  Baseline score:100%, Worst Postbaseline score:90% | 3 | 0 | 0 | 0 | 1 | 1 | 1 | 0
  Baseline score: 70%, Worst Postbaseline score: 60% | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Baseline score: 80%, Worst Postbaseline score: 60% | 0 | 1 | 1 | 0 | 1 | 1 | 0 | 0
  Baseline score: 100%, Worst Postbaseline score:60% | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Baseline score: 80%, Worst Postbaseline score: 70% | 0 | 1 | 0 | 0 | 0 | 0 | 3 | 0
  Baseline score: 90%, Worst Postbaseline score: 70% | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
  Baseline score: 90%, Worst Postbaseline score: 80% | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0
  Baseline score:100%, Worst Postbaseline score:100% | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 5
  Baseline score: 80%, Worst Postbaseline score: 40% | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Baseline score: 70%, Worst Postbaseline score: 80% | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
  Baseline score: 80%, Worst Postbaseline score: 80% | 0 | 0 | 1 | 0 | 2 | 2 | 0 | 2
  Baseline score: 100%, Worst Postbaseline score:80% | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
  Baseline score: 90%, Worst Postbaseline score: 90% | 0 | 0 | 0 | 0 | 4 | 0 | 1 | 2
  Baseline score: 60%, Worst Postbaseline score: 60% | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
  Baseline score: 90%, Worst Postbaseline score: 60% | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Baseline score: 70%, Worst Postbaseline score: 70% | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
  Baseline score: 90%, Worst Postbaseline score:100% | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Baseline score: 100%, Worst Postbaseline score:70% | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Baseline score: 80%, Worst Postbaseline score: 50% | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0

17. Secondary Outcome: Cohorts 1, 2A, 2B, 3A and 3B: Number of Participants With Shift From Baseline to Worst Post Baseline Score in Karnofsky Performance Status (KPS) Scores
Description: KPS: compare effectiveness of medicine for disease and assess outcomes in participants. KPS Scores: recorded on 11 point scale (0, 10, 20, 30, 40, 50, 60, 70, 80, 90 and 100%), where 0=Dead; 10=moribund, fatal processes progressing rapidly; 20=very sick, hospital admission necessary, active supportive treatment necessary; 30=severely disabled, hospital admission is indicated although death not imminent; 40=disabled, requires special care/assistance; 50=requires considerable assistance/frequent medical care; 60=requires occasional assistance, but is able to care for personal needs; 70=cares for self, unable to carry normal activity or active work; 80=normal activity with effort, some signs of disease; 90=able to carry on normal activity, minor signs of disease; 100=normal no complaints, no evidence of disease. Lower score, worse survival for most serious illnesses.
Time Frame: Baseline up to approximately 4 years 7 months
Population: as for outcome 15
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1, Single-agent Dose-finding: Lenvatinib 11 mg/m^2 | Cohort 1, Single-agent Dose-finding: Lenvatinib 14 mg/m^2 | Cohort 1, Single-agent Dose-finding: Lenvatinib 17 mg/m^2 | Cohort 2A, Single-agent Expansion, DTC: Lenvatinib 14 mg/m^2 | Cohort2B,Single-agentExpansion,Osteosarcoma:Lenvatinib14mg/m^2 | Cohort 3A, Combination Dose-finding: Lenvatinib 11 mg/m^2 | Cohort 3A, Combination Dose-finding: Lenvatinib 14 mg/m^2 | Cohort 3B, Combination Expansion: Lenvatinib 14 mg/m^2
Number analyzed (Participants) | 1 | 1 | 0 | 1 | 12 | 3 | 1 | 9
Participants
  Baseline score: 100%, Worst Postbaseline score:80% | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 2
  Baseline score: 100%, Worst Postbaseline score:90% | 0 | 1 | 0 | 0 | 2 | 1 | 0 | 2
  Baseline score: 70%, Worst Postbaseline score: 70% | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
  Baseline score: 90%, Worst Postbaseline score: 70% | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Baseline score: 80%, Worst Postbaseline score: 80% | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Baseline score: 90%, Worst Postbaseline score: 60% | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Baseline score:100%, Worst Postbaseline score:100% | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 1
  Baseline score: 100%, Worst Postbaseline score:70% | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
  Baseline score: 90%, Worst Postbaseline score: 80% | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Baseline score: 90%, Worst Postbaseline score: 90% | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 1

18. Secondary Outcome: Cohorts 1, 2A, 2B, 3A, and 3B: Plasma Concentrations of Lenvatinib
Description: Duration of each cycle for Cohorts 1, 2A, 2B is 28 days. Duration of each cycle for Cohorts 3A, 3B is 21 days.
Time Frame: Cohorts 1, 2A, 2B: Cycle(C)1 Day(D)1: 0.5-4 hours (h), 6-10 h post-dose, C1D15: pre-dose, 0.5-4 h, 6-10 h post-dose, C2D1: pre-dose, 2-12 h post-dose; Cohorts 3A, 3B: C1D1: 0.5-4 h, 6-10 h post-dose, C2D1: pre-dose, 2-12 h post-dose
Population: Pharmacokinetic (PK) Analysis Set included all participants who had received any study drug and had evaluable PK data. Here "number analyzed, n" signifies participants who were evaluable for this outcome measure at given time points.
Measure: Mean (Standard Deviation); unit: nanogram per milliliter (ng/mL)
Arm/Group | Cohort 1, Single-agent Dose-finding: Lenvatinib 11 mg/m^2 | Cohort 1, Single-agent Dose-finding: Lenvatinib 14 mg/m^2 | Cohort 1, Single-agent Dose-finding: Lenvatinib 17 mg/m^2 | Cohort 2A, Single-agent Expansion, DTC: Lenvatinib 14 mg/m^2 | Cohort2B,Single-agentExpansion,Osteosarcoma:Lenvatinib14mg/m^2 | Cohort 3A, Combination Dose-finding: Lenvatinib 11 mg/m^2 | Cohort 3A, Combination Dose-finding: Lenvatinib 14 mg/m^2 | Cohort 3B, Combination Expansion: Lenvatinib 14 mg/m^2
Number analyzed (Participants) | 5 | 11 | 7 | 1 | 31 | 11 | 11 | 20
nanogram per milliliter (ng/mL)
  Cycle 1 Day 1: 0.5-4 hours: number analyzed (Participants) | 5 | 11 | 7 | 1 | 29 | 11 | 11 | 20
  Cycle 1 Day 1: 0.5-4 hours | 295.6 (214.01) | 134.8 (145.83) | 52.5 (81.40) | 11.1 (NA) — Standard deviation could not be calculated because only one participant was available for analysis. | 177.4 (191.03) | 105.2 (131.54) | 111.4 (131.47) | 209.7 (197.66)
  Cycle 1 Day 1: 6-10 hours: number analyzed (Participants) | 5 | 11 | 7 | 1 | 30 | 11 | 11 | 20
  Cycle 1 Day 1: 6-10 hours | 212.7 (185.98) | 281.9 (137.39) | 238.0 (135.87) | 188 (NA) — Standard deviation could not be calculated because only one participant was available for analysis. | 289.4 (200.09) | 191.9 (100.69) | 148.5 (122.41) | 164.8 (73.59)
  Cycle 1 Day 15: Pre-dose: number analyzed (Participants) | 4 | 9 | 6 | 1 | 29 | 0 | 0 | 0
  Cycle 1 Day 15: Pre-dose | 46.9 (11.01) | 59.1 (29.19) | 96.9 (66.10) | 56.2 (NA) — Standard deviation could not be calculated because only one participant was available for analysis. | 67.0 (53.78) |  |  |
  Cycle 1 Day 15: 0.5-4 hours: number analyzed (Participants) | 4 | 8 | 6 | 1 | 28 | 0 | 0 | 0
  Cycle 1 Day 15: 0.5-4 hours | 133.4 (163.37) | 226.6 (204.61) | 191.8 (190.22) | 124 (NA) — Standard deviation could not be calculated because only one participant was available for analysis. | 168.3 (157.67) |  |  |
  Cycle 1 Day 15: 6-10 hours: number analyzed (Participants) | 4 | 8 | 6 | 1 | 29 | 0 | 0 | 0
  Cycle 1 Day 15: 6-10 hours | 351.8 (157.15) | 375.8 (121.21) | 413.0 (221.47) | 247 (NA) — Standard deviation could not be calculated because only one participant was available for analysis. | 322.9 (138.87) |  |  |
  Cycle 2 Day 1: Pre-dose: number analyzed (Participants) | 5 | 8 | 7 | 1 | 27 | 11 | 8 | 17
  Cycle 2 Day 1: Pre-dose | 58.1 (19.58) | 61.6 (60.61) | 97.9 (77.08) | 59.8 (NA) — Standard deviation could not be calculated because only one participant was available for analysis. | 66.8 (62.50) | 51.7 (44.23) | 76.1 (63.25) | 50.4 (65.10)
  Cycle 2 Day 1: 2-12 hours: number analyzed (Participants) | 5 | 7 | 7 | 1 | 28 | 11 | 9 | 18
  Cycle 2 Day 1: 2-12 hours | 502.4 (360.71) | 440.7 (229.29) | 339.2 (212.44) | 102 (NA) — Standard deviation could not be calculated because only one participant was available for analysis. | 382.4 (217.49) | 205.6 (134.66) | 237.4 (124.82) | 275.3 (135.73)

19. Secondary Outcome: Cohort 2B, 3B: Percent Change From Baseline in Serum Biomarkers Level
Description: Serum biomarkers included Fibroblast Growth Factor (FGF) 19, FGF 21, Vascular Endothelial Growth Factor (VEGF). In this outcome measure, percent change from baseline in serum biomarkers level per "PFS-4, Yes" and "PFS-4, No" have been reported. As per assessment of investigator based on RECIST v1.1, "PFS-4, Yes"= participants evaluable for PFS-4 month and alive and without PD at 4 months from the first dose, "PFS-4, No"=participants evaluable for PFS-4 month and not alive or with PD at 4 months from the first dose.
Time Frame: Cohort 2B: Baseline, Cycle 2-3 Day 1 (Duration of each cycle=28 days); Cohort 3B: Baseline, Cycle 2 Day 1, Cycle 4 Day 1 (Duration of each cycle=21 days)
Population: PFS-4 evaluable set: all participants treated with study drug for at least 4 months or those who died or radiologically progressed within 4 months after first dose or received anticancer treatment within 4 months after first dose. "N": participants evaluable for this measure. "n": participants who were evaluable for this measure for specific rows.
Measure: Mean (Standard Deviation); unit: percent change
Groups:
- Cohort2B,Single-agentExpansion,Osteosarcoma:Lenvatinib14mg/m^2: Participants with relapsed or refractory osteosarcoma received lenvatinib 14 mg/m^2 (administered per BSA with daily dose capped at 24 mg/day) as capsule or suspension (lenvatinib capsules were dissolved in water or apple juice for participants who were unable to swallow capsules and given as suspension), orally, once daily on Days 1 to 28 of each treatment cycle as a single agent until PD, intolerable toxicity, participant noncompliance with safety or efficacy assessments, initiation of another anticancer therapy, voluntary discontinuation by the participant at any time, or study termination by the sponsor, whichever occurred first. Duration of each treatment cycle=28 days.
- Cohort 3B, Combination Expansion: Lenvatinib 14 mg/m^2: Participants with relapsed or refractory osteosarcoma received lenvatinib 14 mg/m^2 (administrated per BSA with daily dose capped at 24 mg/day) as capsules or suspension (lenvatinib capsules were dissolved in water or apple juice for participants who were unable to swallow capsules and given as suspension), orally, once daily on Days 1 to 21 of each treatment cycle in combination with ifosfamide 3000 mg/m^2/day intravenously and etoposide 100 mg/m^2/day intravenously on Days 1 to 3 of each treatment cycle for up to a total of 5 cycles as a combination therapy. Duration of each treatment cycle=21 days.
Arm/Group | Cohort2B,Single-agentExpansion,Osteosarcoma:Lenvatinib14mg/m^2 | Cohort 3B, Combination Expansion: Lenvatinib 14 mg/m^2
Number analyzed (Participants) | 26 | 13
percent change
  C2D1: FGF 19 (PFS-4, Yes): number analyzed (Participants) | 8 | 9
  C2D1: FGF 19 (PFS-4, Yes) | 48.7 (110.78) | 172.1 (211.86)
  C2D1: FGF 19 (PFS-4, No): number analyzed (Participants) | 18 | 4
  C2D1: FGF 19 (PFS-4, No) | 109.9 (139.19) | 78.3 (203.30)
  C3D1: FGF 19 (PFS-4, Yes): number analyzed (Participants) | 9 | 0
  C3D1: FGF 19 (PFS-4, Yes) | 47.3 (130.42) |
  C3D1: FGF 19 (PFS-4, No): number analyzed (Participants) | 8 | 0
  C3D1: FGF 19 (PFS-4, No) | 194.5 (180.71) |
  C4D1: FGF 19 (PFS-4, Yes): number analyzed (Participants) | 0 | 9
  C4D1: FGF 19 (PFS-4, Yes) |  | 237.7 (204.94)
  C4D1: FGF 19 (PFS-4, No): number analyzed (Participants) | 0 | 1
  C4D1: FGF 19 (PFS-4, No) |  | 91.9 (NA) — Standard deviation could not be estimated as insufficient number of participants were available for analysis.
  C2D1: FGF 21 (PFS-4, Yes): number analyzed (Participants) | 8 | 9
  C2D1: FGF 21 (PFS-4, Yes) | -14.9 (68.95) | 70.2 (138.90)
  C2D1: FGF 21 (PFS-4, No): number analyzed (Participants) | 18 | 4
  C2D1: FGF 21 (PFS-4, No) | 134.3 (203.81) | 7.2 (48.64)
  C3D1: FGF 21 (PFS-4, Yes): number analyzed (Participants) | 9 | 0
  C3D1: FGF 21 (PFS-4, Yes) | 55.0 (125.51) |
  C3D1: FGF 21 (PFS-4, No): number analyzed (Participants) | 8 | 0
  C3D1: FGF 21 (PFS-4, No) | 17.0 (88.92) |
  C4D1: FGF 21 (PFS-4, Yes): number analyzed (Participants) | 0 | 9
  C4D1: FGF 21 (PFS-4, Yes) |  | 256.2 (323.34)
  C4D1: FGF 21 (PFS-4, No): number analyzed (Participants) | 0 | 1
  C4D1: FGF 21 (PFS-4, No) |  | -1.5 (NA) — Standard deviation could not be estimated as insufficient number of participants were available for analysis.
  C2D1: VEGF (PFS-4, Yes): number analyzed (Participants) | 7 | 9
  C2D1: VEGF (PFS-4, Yes) | 119.9 (309.01) | 87.9 (105.60)
  C2D1: VEGF (PFS-4, No): number analyzed (Participants) | 18 | 4
  C2D1: VEGF (PFS-4, No) | 124.2 (212.18) | 95.8 (92.53)
  C3D1: VEGF (PFS-4, Yes): number analyzed (Participants) | 8 | 0
  C3D1: VEGF (PFS-4, Yes) | 64.3 (153.50) |
  C3D1: VEGF (PFS-4, No): number analyzed (Participants) | 8 | 0
  C3D1: VEGF (PFS-4, No) | 23.2 (69.67) |
  C4D1: VEGF (PFS-4, Yes): number analyzed (Participants) | 0 | 9
  C4D1: VEGF (PFS-4, Yes) |  | 84.3 (97.85)
  C4D1: VEGF (PFS-4, No): number analyzed (Participants) | 0 | 0
Statistical Analysis 1: Comparison: Cohort2B,Single-agentExpansion,Osteosarcoma:Lenvatinib14mg/m^2; C2D1: FGF 19 (PFS-4, Yes) vs. C2D1: FGF 19 (PFS-4, No); Test type: Other; p = 0.20359, Wilcoxon Rank-Sum Test
Statistical Analysis 2: Comparison: Cohort 3B, Combination Expansion: Lenvatinib 14 mg/m^2; C2D1: FGF 19 (PFS-4, Yes) vs. C2D1: FGF 19 (PFS-4, No); Test type: Other; p = 0.50068, Wilcoxon Rank-Sum Test
Statistical Analysis 3: Comparison: Cohort2B,Single-agentExpansion,Osteosarcoma:Lenvatinib14mg/m^2; C3D1: FGF 19 (PFS-4, Yes) vs. C3D1: FGF 19 (PFS-4, No); Test type: Other; p = 0.05512, Wilcoxon Rank-Sum Test
Statistical Analysis 4: Comparison: Cohort 3B, Combination Expansion: Lenvatinib 14 mg/m^2; C4D1: FGF 19 (PFS-4, Yes) vs. C4D1: FGF 19 (PFS-4, No); Test type: Other; p = 0.50382, Wilcoxon Rank-Sum Test
Statistical Analysis 5: Comparison: Cohort2B,Single-agentExpansion,Osteosarcoma:Lenvatinib14mg/m^2; C2D1: FGF 21 (PFS-4, Yes) vs. C2D1: FGF 21 (PFS-4, No); Test type: Other; p = 0.04760, Wilcoxon Rank-Sum Test
Statistical Analysis 6: Comparison: Cohort 3B, Combination Expansion: Lenvatinib 14 mg/m^2; C2D1: FGF 21 (PFS-4, Yes) vs. C2D1: FGF 21 (PFS-4, No); Test type: Other; p = 0.21420, Wilcoxon Rank-Sum Test
Statistical Analysis 7: Comparison: Cohort2B,Single-agentExpansion,Osteosarcoma:Lenvatinib14mg/m^2; C3D1: FGF 21 (PFS-4, Yes) vs. C3D1: FGF 21 (PFS-4, No); Test type: Other; p = 0.42542, Wilcoxon Rank-Sum Test
Statistical Analysis 8: Comparison: Cohort 3B, Combination Expansion: Lenvatinib 14 mg/m^2; C4D1: FGF 21 (PFS-4, Yes) vs. C4D1: FGF 21 (PFS-4, No); Test type: Other; p = 0.73573, Wilcoxon Rank-Sum Test
Statistical Analysis 9: Comparison: Cohort2B,Single-agentExpansion,Osteosarcoma:Lenvatinib14mg/m^2; C2D1: VEGF (PFS-4, Yes) vs. C2D1: VEGF (PFS-4, No); Test type: Other; p = 0.35754, Wilcoxon Rank-Sum Test
Statistical Analysis 10: Comparison: Cohort 3B, Combination Expansion: Lenvatinib 14 mg/m^2; C2D1: VEGF (PFS-4, Yes) vs. C2D1: VEGF (PFS-4, No); Test type: Other; p = 0.59903, Wilcoxon Rank-Sum Test
Statistical Analysis 11: Comparison: Cohort2B,Single-agentExpansion,Osteosarcoma:Lenvatinib14mg/m^2; C3D1: VEGF (PFS-4, Yes) vs. C3D1: VEGF (PFS-4, No); Test type: Other; p = 1.00000, Wilcoxon Rank-Sum Test

20. Secondary Outcome: Cohorts 1, 2A, 2B, 3A and 3B: Number of Participants With Most Frequent Treatment-emergent Adverse Events (TEAEs) Related to Lenvatinib Exposure
Description: TEAEs (serious and non-serious), those occurred most frequently have been reported in this outcome measure. "Palmar-plantar E syndrome" refers to Palmar-plantar erythrodysaesthesia syndrome.
Time Frame: First dose of study drug until 30 days after last dose of study drug (Cohort 1, Cohort 2A, Cohort 2B: until the data cut-off date, 31 May 2019; Cohort 3A, Cohort 3B: until the data cut-off date, 18 July 2019)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1, Single-agent Dose-finding: Lenvatinib 11 mg/m^2 | Cohort 1, Single-agent Dose-finding: Lenvatinib 14 mg/m^2 | Cohort 1, Single-agent Dose-finding: Lenvatinib 17 mg/m^2 | Cohort 2A, Single-agent Expansion, DTC: Lenvatinib 14 mg/m^2 | Cohort2B,Single-agentExpansion,Osteosarcoma:Lenvatinib14mg/m^2 | Cohort 3A, Combination Dose-finding: Lenvatinib 11 mg/m^2 | Cohort 3A, Combination Dose-finding: Lenvatinib 14 mg/m^2 | Cohort 3B, Combination Expansion: Lenvatinib 14 mg/m^2
Number analyzed (Participants) | 5 | 11 | 7 | 1 | 31 | 11 | 11 | 20
Participants
  Hypothyroidism | 3 | 6 | 3 | 0 | 13 | 5 | 6 | 6
  Abdominal pain | 2 | 2 | 1 | 1 | 5 | 6 | 5 | 6
  Diarrhea | 3 | 5 | 3 | 1 | 8 | 5 | 5 | 12
  Nausea | 1 | 2 | 3 | 0 | 8 | 7 | 8 | 13
  Vomiting | 1 | 6 | 3 | 0 | 7 | 5 | 6 | 12
  Asthenia | 2 | 1 | 0 | 0 | 8 | 0 | 0 | 7
  Fatigue | 2 | 2 | 3 | 0 | 8 | 2 | 4 | 3
  Alanine aminotransferase increased | 0 | 2 | 1 | 0 | 1 | 3 | 1 | 4
  Blood thyroid stimulating hormone increased | 0 | 0 | 0 | 0 | 9 | 3 | 0 | 5
  Weight decreased | 3 | 4 | 1 | 0 | 6 | 5 | 3 | 4
  Decreased appetite | 3 | 5 | 1 | 0 | 13 | 4 | 2 | 5
  Arthralgia | 0 | 2 | 1 | 0 | 1 | 2 | 4 | 1
  Myalgia | 1 | 2 | 0 | 0 | 1 | 0 | 0 | 0
  Pain in extremity | 0 | 2 | 1 | 0 | 0 | 3 | 1 | 0
  Headache | 0 | 1 | 1 | 0 | 5 | 2 | 4 | 4
  Proteinuria | 0 | 3 | 3 | 0 | 7 | 2 | 5 | 8
  Dysphonia | 0 | 0 | 0 | 0 | 5 | 0 | 0 | 0
  Erythema | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0
  Hair color changes | 1 | 1 | 1 | 0 | 2 | 0 | 0 | 0
  Palmar-plantar E syndrome | 2 | 2 | 0 | 0 | 1 | 1 | 2 | 0
  Hypertension | 2 | 3 | 4 | 1 | 10 | 1 | 4 | 3
  Haematuria | 0 | 0 | 0 | 0 | 0 | 4 | 1 | 4
  Hypokalaemia | 0 | 0 | 0 | 0 | 0 | 4 | 1 | 2
  Hypophosphataemia | 0 | 0 | 0 | 0 | 0 | 3 | 2 | 2
  Platelet count decreased | 0 | 0 | 0 | 0 | 0 | 2 | 3 | 11
  Back pain | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 2
  Dry skin | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 0
  Oral pain | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 1
  Pneumothorax | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 1
  Dehydration | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 4
  Hypoalbuminaemia | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0
  Lethargy | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 2
  Leukopenia | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 3
  Neutrophil count decreased | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 9
  Oral dysaesthesia | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0
  Oropharyngeal pain | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 1
  Proctalgia | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0
  Toxic encephalopathy | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0
  Lymphocyte count decreased | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 4
  Abdominal pain upper | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 4
  Hyperuricemia | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Insomnia | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Anaemia | 0 | 0 | 0 | 0 | 0 | 9 | 7 | 15
  Neutropenia | 0 | 0 | 0 | 0 | 0 | 6 | 6 | 8
  Epistaxis | 0 | 0 | 0 | 0 | 0 | 5 | 4 | 4
  Thrombocytopenia | 0 | 0 | 0 | 0 | 0 | 5 | 4 | 5
  Febrile neutropenia | 0 | 0 | 0 | 0 | 0 | 5 | 3 | 2
  Stomatitis | 0 | 0 | 0 | 0 | 0 | 4 | 4 | 4
  Constipation | 0 | 0 | 0 | 0 | 0 | 5 | 2 | 2
  White blood cell count decreased | 0 | 0 | 0 | 0 | 0 | 4 | 3 | 12
  Lymphopenia | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
  Haematochezia | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
  Pyrexia | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
  Wound dehiscence | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
  Hypocalcaemia | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
  Dizziness | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
  Dyspnoea | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
  Hyperhidrosis | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0

21. Secondary Outcome: Cohorts 1, 2A, 2B, 3A and 3B: Number of Participants Categorized Based on Overall Acceptability Questionnaire Responses for Suspension of Lenvatinib
Description: In acceptability questionnaire, participants were asked to answer the overall acceptability of lenvatinib suspension considering the following elements: taste, appearance, smell and how does it feel in the mouth. Overall acceptability was answered in terms of 7 responses: Super good, really good, good, may be good or may be bad, bad, really bad, super bad. Overall acceptability was the overall acceptance for taste, appearance, smell, and the feeling in mouth. In this measure, number of participants have been reported per their overall acceptability responses.
Time Frame: Cycle 1 Day 1 (Cycle length=28 days for Cohorts 1, 2A, 2B; Cycle length=21 days for Cohorts 3A, 3B)
Population: Palatability analysis set included all participants who received oral suspension of lenvatinib and answered at least 1 question in the palatability questionnaire case report form.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1, Single-agent Dose-finding: Lenvatinib 11 mg/m^2 | Cohort 1, Single-agent Dose-finding: Lenvatinib 14 mg/m^2 | Cohort 1, Single-agent Dose-finding: Lenvatinib 17 mg/m^2 | Cohort 2A, Single-agent Expansion, DTC: Lenvatinib 14 mg/m^2 | Cohort2B,Single-agentExpansion,Osteosarcoma:Lenvatinib14mg/m^2 | Cohort 3A, Combination Dose-finding: Lenvatinib 11 mg/m^2 | Cohort 3A, Combination Dose-finding: Lenvatinib 14 mg/m^2 | Cohort 3B, Combination Expansion: Lenvatinib 14 mg/m^2
Number analyzed (Participants) | 0 | 2 | 1 | 0 | 1 | 0 | 1 | 4
Participants
  Super Good | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Really Good | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Good | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 1
  May be Good or May be Bad | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Bad | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Really Bad | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
  Super Bad | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: From the date of first dose of study drug up to 30 days after the last dose (up to approximately 7 years)
Description: Safety analysis set included all participants who received any study drug and had at least one post-baseline safety evaluation. The difference in the numbers of deaths in the Participant Flow module versus the Adverse Events module is because the deaths presented in the Participant Flow module are based from the Full Analysis Set while the deaths presented in the Adverse Events module are based from the Safety Population.
Groups:
- Lenvatinib 5 mg/m^2: Eligible participants of age group 2 to <6 years first underwent a 21-day run-in period with lenvatinib 5 mg/m^2, once daily as capsule or suspension (lenvatinib capsules were dissolved in water or apple juice for participants who were unable to swallow capsules and given as suspension) before receiving lenvatinib 11 mg/m^2 or 14 mg/m^2 in Cycle 1 of Cohort 1 (Single-agent Dose-finding).
Arm/Group | Lenvatinib 5 mg/m^2 | Cohort 1, Single-agent Dose-finding: Lenvatinib 11 mg/m^2 | Cohort 1, Single-agent Dose-finding: Lenvatinib 14 mg/m^2 | Cohort 1, Single-agent Dose-finding: Lenvatinib 17 mg/m^2 | Cohort 2A, Single-agent Expansion, DTC: Lenvatinib 14 mg/m^2 | Cohort2B,Single-agentExpansion,Osteosarcoma:Lenvatinib14mg/m^2 | Cohort 3A, Combination Dose-finding: Lenvatinib 11 mg/m^2 | Cohort 3A, Combination Dose-finding: Lenvatinib 14 mg/m^2 | Cohort 3B, Combination Expansion: Lenvatinib 14 mg/m^2
All-Cause Mortality (participants affected / at risk) | 0/2 | 2/5 | 7/11 | 6/7 | 0/1 | 27/31 | 10/11 | 6/11 | 14/20
Serious Adverse Events (participants affected / at risk) | 0/2 | 3/5 | 7/11 | 5/7 | 1/1 | 21/31 | 7/11 | 9/11 | 16/20
Other Adverse Events (participants affected / at risk) | 2/2 | 5/5 | 11/11 | 7/7 | 1/1 | 29/31 | 11/11 | 11/11 | 20/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lenvatinib 5 mg/m^2 (N=2) | Cohort 1, Single-agent Dose-finding: Lenvatinib 11 mg/m^2 (N=5) | Cohort 1, Single-agent Dose-finding: Lenvatinib 14 mg/m^2 (N=11) | Cohort 1, Single-agent Dose-finding: Lenvatinib 17 mg/m^2 (N=7) | Cohort 2A, Single-agent Expansion, DTC: Lenvatinib 14 mg/m^2 (N=1) | Cohort2B,Single-agentExpansion,Osteosarcoma:Lenvatinib14mg/m^2 (N=31) | Cohort 3A, Combination Dose-finding: Lenvatinib 11 mg/m^2 (N=11) | Cohort 3A, Combination Dose-finding: Lenvatinib 14 mg/m^2 (N=11) | Cohort 3B, Combination Expansion: Lenvatinib 14 mg/m^2 (N=20)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (5)
Cardiac arrest (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardio-respiratory arrest (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Enterocolitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 2 (4)
Gait disturbance (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
General physical health deterioration (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Amylase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood pressure increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ejection fraction decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lipase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (5) | 0 (0) | 0 (0) | 4 (12)
Weight decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 4 (4) | 1 (1) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depressed level of consciousness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spinal cord compression (Nervous system disorders) | 0 (0) | 0 (0) | 1 (4) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 1 (1)
Gingival bleeding (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1)
Facial pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 2 (2)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Wound dehiscence (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Intervertebral disc compression (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 1 (4)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Renal pain (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (2) | 0 (0) | 1 (2)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (5) | 0 (0) | 0 (0) | 0 (0) | 4 (7) | 2 (3) | 2 (2) | 3 (4)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Arterial thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lymphoedema (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (8) | 3 (4) | 2 (5)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Clostridium difficile infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Wound infection bacterial (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Accidental overdose (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Brain injury (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Toxic encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 1 (1)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pancytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cardiac failure (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anal inflammation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vulvitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Allergic transfusion reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Transfusion related complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (18)
White blood cell count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (16)
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Renal failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Venoocclusive disease (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dysmetria (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Suicide attempt (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lenvatinib 5 mg/m^2 (N=2) | Cohort 1, Single-agent Dose-finding: Lenvatinib 11 mg/m^2 (N=5) | Cohort 1, Single-agent Dose-finding: Lenvatinib 14 mg/m^2 (N=11) | Cohort 1, Single-agent Dose-finding: Lenvatinib 17 mg/m^2 (N=7) | Cohort 2A, Single-agent Expansion, DTC: Lenvatinib 14 mg/m^2 (N=1) | Cohort2B,Single-agentExpansion,Osteosarcoma:Lenvatinib14mg/m^2 (N=31) | Cohort 3A, Combination Dose-finding: Lenvatinib 11 mg/m^2 (N=11) | Cohort 3A, Combination Dose-finding: Lenvatinib 14 mg/m^2 (N=11) | Cohort 3B, Combination Expansion: Lenvatinib 14 mg/m^2 (N=20)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (2) | 2 (2) | 1 (1) | 0 (0) | 5 (7) | 9 (43) | 7 (29) | 15 (77)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (4) | 0 (0) | 0 (0) | 2 (8) | 0 (0) | 2 (3)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 6 (19) | 6 (25) | 8 (51)
Polycythaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 3 (7) | 5 (50) | 4 (54) | 5 (47)
Pericardial effusion (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 2 (2)
Hypothyroidism (Endocrine disorders) | 1 (1) | 3 (5) | 6 (10) | 3 (3) | 0 (0) | 13 (17) | 6 (7) | 8 (11) | 6 (8)
Eye ulcer (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Papilloedema (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 2 (3) | 7 (9) | 2 (6) | 1 (1) | 9 (27) | 6 (20) | 6 (18) | 7 (23)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 4 (9) | 0 (0) | 1 (1) | 4 (8)
Anal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anal incontinence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anal pruritus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aphthous ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 10 (14) | 6 (11) | 5 (8) | 7 (10)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 4 (5) | 5 (9) | 4 (8) | 1 (12) | 12 (29) | 8 (24) | 6 (14) | 13 (72)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 5 (5) | 0 (0) | 0 (0) | 4 (7)
Flatulence (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Gingival pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mouth ulceration (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 3 (8) | 2 (4) | 3 (3) | 0 (0) | 12 (16) | 8 (28) | 8 (28) | 14 (45)
Odynophagia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 2 (2) | 2 (2)
Oral dysaesthesia (Gastrointestinal disorders) | 0 (0) | 1 (2) | 1 (6) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 1 (1) | 0 (0)
Perianal erythema (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Proctalgia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 3 (5) | 2 (2) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 2 (3)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 4 (5) | 5 (7) | 3 (4) | 4 (8)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (9) | 7 (20) | 4 (5) | 0 (0) | 14 (41) | 9 (28) | 8 (20) | 12 (58)
Asthenia (General disorders) | 0 (0) | 2 (4) | 1 (1) | 0 (0) | 0 (0) | 10 (13) | 1 (9) | 2 (3) | 8 (28)
Catheter site pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1)
Fatigue (General disorders) | 1 (1) | 2 (4) | 3 (4) | 3 (7) | 0 (0) | 9 (15) | 4 (8) | 6 (9) | 4 (4)
Non-cardiac chest pain (General disorders) | 0 (0) | 2 (6) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 3 (4) | 1 (3)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 1 (1) | 1 (5) | 1 (1) | 0 (0) | 4 (4) | 1 (1) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 2 (8) | 4 (9) | 4 (10) | 1 (1) | 11 (17) | 6 (6) | 3 (5) | 6 (9)
Hepatocellular injury (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Ear infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Localised infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0)
Oral candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Rhinitis (Infections and infestations) | 2 (2) | 1 (2) | 2 (3) | 3 (3) | 0 (0) | 4 (4) | 1 (1) | 1 (1) | 2 (2)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Staphylococcal sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (4) | 1 (1) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (2) | 1 (1) | 1 (3) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 2 (2)
Viral infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vulvovaginal candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 4 (6) | 2 (4) | 1 (1) | 1 (1) | 3 (3) | 1 (2) | 5 (13)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 3 (3) | 2 (6) | 1 (1) | 2 (2) | 1 (1) | 1 (3) | 3 (13)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 3 (4) | 1 (1) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 2 (3)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 1 (1)
Blood lactate dehydrogenase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Blood urea increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
C-reactive protein increased (Investigations) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 2 (2)
Ejection fraction decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (2) | 1 (1) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 2 (5) | 1 (1) | 1 (4) | 2 (4)
Lipase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 2 (2)
Neutrophil count increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 2 (14) | 2 (12) | 4 (16) | 11 (86)
Red blood cell sedimentation rate increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 3 (13) | 3 (6) | 3 (5) | 0 (0) | 11 (17) | 6 (8) | 3 (7) | 5 (9)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 4 (14) | 5 (9) | 3 (5) | 0 (0) | 15 (26) | 5 (8) | 3 (3) | 7 (12)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (4) | 0 (0) | 0 (0) | 1 (2) | 2 (4) | 1 (1) | 2 (5)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (2) | 4 (8) | 1 (4) | 3 (10)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 2 (4) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 3 (3) | 1 (1) | 1 (1) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (2) | 0 (0) | 10 (17) | 6 (7) | 6 (8) | 3 (8)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 4 (8) | 2 (2) | 1 (2) | 10 (15) | 6 (7) | 4 (6) | 5 (5)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 6 (6) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (2) | 0 (0) | 10 (14) | 2 (3) | 1 (1) | 3 (5)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (12) | 2 (2) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 2 (3) | 2 (3)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (4) | 4 (10) | 3 (5) | 0 (0) | 9 (10) | 6 (16) | 5 (11) | 3 (4)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2) | 1 (2) | 0 (0) | 0 (0) | 3 (5) | 1 (1) | 0 (0) | 1 (1)
Pericardial effusion malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (4) | 0 (0) | 0 (0) | 0 (0)
Cranial nerve paralysis (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 3 (3) | 1 (1) | 3 (5) | 2 (2)
Dysaesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (2) | 6 (9) | 3 (6) | 0 (0) | 15 (20) | 4 (5) | 7 (13) | 6 (10)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Lethargy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 1 (1) | 2 (2)
Monoparesis (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle contractions involuntary (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Phantom pain (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pyramidal tract syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sciatica (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 3 (3) | 3 (8) | 1 (1) | 2 (2)
Depressed mood (Psychiatric disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Sleep disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Bladder pain (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cystitis noninfective (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 2 (3) | 1 (3)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 2 (2) | 5 (6) | 1 (2) | 4 (12)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Proteinuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 3 (16) | 3 (8) | 0 (0) | 13 (27) | 3 (5) | 5 (13) | 9 (44)
Menstruation irregular (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (3) | 3 (3) | 2 (2) | 0 (0) | 9 (10) | 4 (4) | 4 (5) | 6 (6)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 6 (10) | 1 (2) | 2 (3) | 1 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (3) | 0 (0) | 1 (2) | 0 (0) | 6 (8) | 3 (3) | 2 (3) | 2 (3)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (3) | 3 (3) | 2 (2) | 1 (1) | 4 (7) | 5 (10) | 6 (8) | 7 (15)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (6) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 1 (1) | 2 (2) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 3 (4) | 3 (3) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0)
Hair colour changes (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Pain of skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (4) | 2 (2) | 0 (0) | 1 (2) | 1 (2) | 1 (1) | 3 (12) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (4) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 2 (3) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 3 (7) | 2 (4)
Rash macular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Rash papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spider naevus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flushing (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 2 (2) | 3 (3) | 4 (12) | 1 (2) | 10 (13) | 3 (4) | 5 (10) | 5 (6)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thyroglobulin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (8) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperuricaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 1 (1) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 3 (7) | 1 (1) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Left ventricular dysfunction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Anal fissure (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (5) | 0 (0) | 2 (2) | 2 (2)
Eructation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (2) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Blood thyroid stimulating hormone increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 9 (13) | 3 (4) | 0 (0) | 5 (8)
Electrocardiogram QT prolonged (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 1 (2)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 2 (3) | 0 (0) | 3 (3)
Neuralgia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (2) | 2 (3)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (5) | 1 (1) | 0 (0) | 0 (0)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (4) | 2 (21) | 3 (20)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 4 (4) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0)
Diplopia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dry eye (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Eye pain (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Eyelid oedema (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (4) | 0 (0) | 0 (0)
Ocular hyperaemia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Photophobia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Anal fistula (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anal inflammation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Anal skin tags (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea haemorrhagic (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (4) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Glossitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 1 (4)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hypoaesthesia oral (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oesophageal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oral discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oral pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 3 (3) | 1 (1)
Proctitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Catheter site bruise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Catheter site dermatitis (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Catheter site swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chills (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Device related thrombosis (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Face oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infusion site irritation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Localised oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Malaise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (10) | 0 (0) | 1 (1) | 0 (0)
Clostridium difficile infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Cystitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Device related infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Eye infection bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gingivitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Oral herpes (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Osteomyelitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Paronychia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Pseudomonas infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash pustular (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (2)
Staphylococcal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Vascular device infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Allergic transfusion reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (6) | 1 (2) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 2 (2)
Wound (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Wound complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Wound dehiscence (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Blood calcium decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood magnesium decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (10) | 0 (0) | 0 (0)
Blood phosphorus increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood potassium decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 2 (5)
Haemoglobin decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 4 (19) | 2 (5) | 6 (15)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (5) | 10 (46)
Thyroxine decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urine output decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
White blood cell count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (8) | 4 (11) | 13 (88)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (4) | 2 (2)
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (4) | 0 (0)
Hypermagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 2 (3) | 0 (0) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (8) | 2 (13) | 4 (12)
Hypoproteinaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Metabolic acidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Coccydynia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Groin pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Periostitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Amputation stump pain (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Generalised tonic-clonic seizure (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Migraine (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (8) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sensory disturbance (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Toxic encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Agitation (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Irritability (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Glycosuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Renal impairment (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Renal tubular disorder (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Balanoposthitis (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vulvovaginal pruritus (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dysaesthesia pharynx (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 4 (4) | 4 (8)
Pharyngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Dermatitis bullous (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Scab (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lymphoedema (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acquired antithrombin III deficiency (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4)
Ventricular dysfunction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (5)
Eye discharge (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyschezia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haematemesis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Noninfective gingivitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Axillary pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Inflammation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Eyelid infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Folliculitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oesophageal candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vaginal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Amylase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Blood phosphorus decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood uric acid decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Culture stool positive (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Full blood count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lipase decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cachexia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fluid retention (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1)
Limb mass (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nightmare (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Leukocyturia (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (9)
Renal failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Urine flow decreased (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Genital pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Onychalgia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash generalised (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Capillary leak syndrome (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haematoma (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hot flush (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (3)
Bundle branch block right (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiotoxicity (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anal fissure haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mouth haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Paraesthesia oral (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Injection site mass (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sensation of foreign body (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anal fungal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Angular cheilitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Catheter site infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Genital candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Genital infection fungal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tonsillitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anaemia postoperative (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Post procedural complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Vaccination complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Brain natriuretic peptide increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Coronavirus test positive (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Electrocardiogram PR prolongation (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Occult blood positive (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1)
Thyroxine increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Weight increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
White blood cell count increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypochloraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperamylasaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle atrophy (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Muscle rigidity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Major depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mood altered (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Albuminuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Nephropathy toxic (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Amenorrhoea (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Genital lesion (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Perineal pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Premature menopause (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (4) | 0 (0) | 0 (0) | 0 (0)
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Itching scar (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Palmar erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Scar pain (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Umbilical discharge (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Purpura (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cardiac dysfunction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Systolic dysfunction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gingival bleeding (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Abscess limb (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Superior vena cava syndrome (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2019-11-22): https://cdn.clinicaltrials.gov/large-docs/74/NCT02432274/Prot_002.pdf
  • Statistical Analysis Plan (2019-03-26): https://cdn.clinicaltrials.gov/large-docs/74/NCT02432274/SAP_003.pdf